CLINICAL TRIAL: NCT03044353
Title: A Multiple Treatment Session, Open Label Phase 2 Clinical Study of GSK2398852 Administered Following and Together With GSK2315698 in Cohorts of Patients With Cardiac Amyloidosis
Brief Title: Multiple Treatment Session Study to Assess GSK2398852 Administered Following and Along With GSK2315698
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in benefit/risk profile
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201464; 2016-000276-23 (EudraCT Number)
Record Dates: First submitted 2016-06-27; First posted 2017-02-07 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: Amyloidosis
Keywords: echocardiography (ECHO); skin biopsy; monoclonal anti-serum amyloid p component antibody (anti-SAP mAb); Amyloidosis; cardiac magnetic resonance imaging (CMR); biomarkers; cardiac functional measures; left ventricular mass
MeSH Terms: conditions — Amyloidosis | interventions — miridesap; dezamizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Cardiac TTR amyloidosis (ATTR-CM) participants (Experimental): Cardiac transthyretin (TTR) amyloidosis (transthyretin amyloid cardiomyopathy [ATTR-CM]) participants with mutant genotypes primarily associated with familial amyloidotic cardiomyopathy (FAC) and wild-type TTR will be included. Participants will receive 6 anti-SAP treatments, consisting of carboxy pyrrolidine hexanoyl pyrrolidine carboxylate (CPHPC) followed by anti-SAP monoclonal antibody (mAb) at monthly intervals. During each anti-SAP treatment, participants will receive CPHPC intravenous (IV) infusion once daily for up to 72 hours. After 72 hours of CPHPC administration, participants will be administered intravenous infusion of anti-SAP mAb over 6-8 hours each on Days 1 and 3. The starting dose level of anti-SAP mAb will be 600 milligrams (mg) (divided into 2 infusions of 300 mg). In each treatment session, CPHPC will be administered as subcutaneous (SC) injection for 11 days from the day of first dose of anti-SAP mAb.
  Interventions: Drug: GSK2315698 (CPHPC); Biological: GSK2398852 (anti-SAP mAb)
- Group 2: Post-chemotherapy AL Amyloidosis participants (Experimental): Immunoglobin light chain amyloidosis (AL) participants who attain either a very good partial response (VGPR), or complete response (CR), to systemic chemotherapy (including autologous stem cell transplantation) will be included. Participants will receive 6 anti-SAP treatments, consisting of CPHPC followed by anti-SAP mAb at monthly intervals. During each anti-SAP treatment, participants will receive CPHPC IV infusion once daily for up to 72 hours. After 72 hours of CPHPC administration, participants will be administered IV infusion of anti-SAP mAb over 6-8 hours each on Days 1 and 3. The starting dose level of anti-SAP mAb will be 600 mg (divided into 2 infusions of 300 mg). In each treatment session, CPHPC will be administered by as SC injection for 11 days from the day of first dose of anti-SAP mAb.
  Interventions: Drug: GSK2315698 (CPHPC); Biological: GSK2398852 (anti-SAP mAb)
- Group 3: Newly diagnosed Mayo stage II/IIIa AL participants (Experimental): Newly diagnosed Mayo stage II/IIIa AL participants who attain a free light chain CR during the first 3 cycles of first-line chemotherapy where the first cycle was cyclophosphamide, bortezomib, dexamethasone (CyBorD) will be included. Participants will receive 6 anti-SAP treatments, consisting of CPHPC followed by anti-SAP mAb at monthly intervals. During each anti-SAP treatment, participants will receive CPHPC IV infusion once daily for up to 72 hours. After 72 hours of CPHPC administration, participants will be administered IV infusion of anti-SAP mAb over 6-8 hours each on Days 1 and 3. The starting dose level of anti-SAP mAb will be 600 mg (divided into 2 infusions of 300 mg). In each treatment session, CPHPC will be administered as SC injection for 11 days from the day of first dose of anti-SAP mAb.
  Interventions: Drug: GSK2315698 (CPHPC); Biological: GSK2398852 (anti-SAP mAb)

INTERVENTIONS:
Drug: GSK2315698 (CPHPC) — 20mg/hour, IV (in the vein) for up to 72hours followed by 60mg three times daily subcutaneous injection for 11 days. Number of cycles: up to 6. Dose level and frequency adjusted according to renal function
Biological: GSK2398852 (anti-SAP mAb) — Up to 1200mg, IV divided over days 1 and 3. Number of cycles: up to 6. Dose level adjusted based on tolerability.

SUMMARY:
The study is intended to evaluate whether monthly repeated courses of administration of GSK2315698 followed by GSK2398852 is associated with a reduction in cardiac amyloid load in patients with cardiac amyloidosis, monitored by cardiac magnetic resonance imaging (CMR) and echocardiography (ECHO), and whether this is associated with an improvement in cardiac function. Cohort 1 is transthyretin cardiomyopathy (ATTR-CM) , cohort 2 is patients with immunoglobulin light chain (AL) systemic amyloidosis at greater than 6 months post chemotherapy, cohort 3 newly diagnosed AL systemic amyloidosis undergoing chemotherapy. Primary objectives for the study are assessment of reduction in cardiac amyloid load after repeated administrations of Anti-SAP treatment as evaluated by CMR in all study groups and assessment of safety & tolerability of repeated administration of Anti-SAP treatment, including compatibility with chemotherapy treatment in patients with AL systemic amyloidosis. This is an open label, non-randomised, three-group, monthly repeat Anti-SAP treatment study in systemic amyloidosis patients with cardiac dysfunction caused by cardiac amyloidosis. Subjects will receive up to 6 courses of Anti-SAP treatment. Maximum total duration for a subject in the study is approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years of age inclusive, at the time of signing the informed consent.
* Male and female.

Males:

Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication for a cycle of spermatogenesis following five terminal half-lives after the last dose of study medication. Vasectomy with documentation of azoospermia.

Male condom plus partner use of one of the contraceptive options below: Contraceptive subdermal implant, Intrauterine device or intrauterine system, Combined Oral Contraceptive or Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches .

This is an all-inclusive list of those methods that meet the following GlaxoSmithKline (GSK) definition of highly effective: having a failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. For non-product methods (e.g., male sterility), the investigator determines what is consistent and correct use. The GSK definition is based on the definition provided by the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH).

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

Females

A female subject is eligible to participate if she is not pregnant (as confirmed by a negative Urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

• Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy.

Postmenopausal defined as: 60 years old; Twelve(12) months of spontaneous amenorrhea with an appropriate clinical profile, e.g. age appropriate, > 45 years, in the absence of hormone replacement therapy (HRT) or medical suppression of the menstrual cycle (e.g. leuprolide treatment) in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and oestradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on HRT and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

• Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) (As mentioned in study protocol) from 30 days prior to the first dose of study medication and until 3 months after the last dose of study medication.

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Late-Gadolinum enhancement (LGE) on CMR indicative of cardiac amyloidosis
* LV mass on CMR > 200 grams (g) Inclusion Criteria for Group 1
* Transthyretin amyloid (ATTR) cardiomyopathy (CM)
* Subjects with a diagnosis of hereditary ATTR amyloidosis should have a known amyloidogenic transthyretin (TTR) mutation demonstrated by genotyping AND is recognised to be primarily associated with cardiomyopathy AND one of the following: Definite histochemical identification of amyloid by Congo red staining and green birefringence in crossed polarised light in cardiac or other tissue biopsy and identification of TTR as the amyloid fibril protein either by immunohistochemistry or proteomic analysis.

Or Scintigraphy: 99m^Tc-DPD with Grade 2 cardiac uptake or 99m^Tc-PYP with either Grade 2 or 3 cardiac uptake.

* Subjects with a diagnosis of wild type ATTR-CM must be negative by genotyping and have one of the following: Definite histochemical identification of amyloid by Congo red staining and green birefringence in crossed polarised light in cardiac or other tissue biopsy and identification of TTR as the amyloid fibril protein either by immunohistochemistry or proteomic analysis OR Scintigraphy 99m^Technetium-dicarboxypropane diphosphonate (99m^Tc-DPD) with Grade 2 cardiac uptake or 99m^ Technetium-pyrophosphate (99m^Tc-PYP) with Grade 2 or 3 cardiac uptake.
* Clinically stable in New York heart association (NYHA) class 2 or 3 for the 3 months preceding screening

Inclusion Criteria for Group 2

* Subject medically diagnosed with AL amyloidosis that has required chemotherapy or an autologous stem cell transplant based upon:

AL amyloidosis confirmed by biopsy with immunohistochemical staining or proteomic identification of AL amyloid fibril type, in subjects with definite monoclonal gammopathy in whom causative mutations of all known relevant amyloidogenic genes have been excluded

* Clinically stable in NYHA class 2 or 3 for the 3 months preceding screening
* >=6 months after completing any line of chemotherapy, or after autologous stem cell transplantation, and having attained either a very good partial response (VGPR) or a complete response (CR), and without the need for haematological maintenance therapies

Inclusion Criteria for Group 3

* Newly diagnosed AL amyloidosis based upon:

AL amyloidosis confirmed by biopsy with immunohistochemical staining or proteomic identification of AL amyloid fibril type in subjects with definite monoclonal gammopathy in whom causative mutations of all known relevant amyloidogenic genes have been excluded

* Mayo stage II or IIIa
* Confirmed free light chain complete response (CR) during the first three cycles of first-line chemotherapy where at least the first cycle has been with cyclophosphamide, bortezomib, dexamethasone (CyBorD).

Exclusion Criteria:

* Cardiomyopathy primarily caused by non-amyloid diseases (e.g. ischemic heart disease; valvular heart disease)
* Interval from the Q wave on the ECG to point T using Fredericia's formula (QTcF) > 500 millisecond (msec)
* Sustained / symptomatic monomorphic ventricular tachycardia (VT), or rapid polymorphic VT, at screening
* Unstable heart failure defined as emergency hospitalization for worsening, or decompensated heart failure, or syncopal episode within 1 month of screening.

Implantable cardiac defibrillator (ICD) or permanent pacemaker (PPM) at screening

* N-terminal pro b-type Natriuretic Peptide [(NT)-proBNP] >8500 nanograms (ng)/ Liter (L)
* Glomerular filtration rate (GFR) at Screening < 40 milliliter (mL)/minute (min)
* Any active and persistent dermatological condition
* Existing diagnosis of any type of dementia
* History of allogeneic stem cell transplantation, prior solid organ transplant, or anticipated to undergo solid organ transplantation, or left ventricular assist device (LVAD) implantation, during the course of the study.
* Malignancy within last 5 years, except for basal or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix that has been successfully treated.
* Acute coronary syndrome, or any form of coronary revascularization procedure (including coronary artery bypass grafting [CABG]), within 6 months of screening.
* Stroke within 6 months of screening, or transient ischaemic attack (TIA) within 3 months of screening
* Symptomatic, clinically significant autonomic neuropathy which the Principal Investigator (PI) feels will preclude administration of study treatment
* Hypoalbuminaemia (serum albumin < 30 g/L)
* Uncontrolled hypertension during screening
* Alanine transaminase ALT >3x upper limit of normal (ULN) AND bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Peripheral oedema at Screening that in the opinion of the Prinicpal Investigator (PI) or designee might prevent adequate absorption of subcutaneously administered CPHPC
* Urine dipstick positive (>1+) for blood during screening with investigation indicating glomerular haematuria. If other causes are identified, subjects may be enrolled on resolution of the abnormality
* Presence of any co-morbid or an uncontrolled medical condition (e.g. diabetes mellitus), which in the opinion of the investigator would increase the potential risk to the subject. Investigator should liaise with the Medical Monitor where there is uncertainty as to the eligibility of a patient
* Positive test for hepatitis B hepatitis C, and / or human immunodeficiency virus (HIV) during screening, or within 3 months prior to first dose of study treatment
* Unwillingness or inability to follow the procedures outlined in the protocol
* Use of GSK2315698 (CPHPC), or participation in a separate clinical trial involving CPHPC within 3 months of screening
* Any prohibited concomitant medication as per protocol within 28 days of Screening
* Donation of blood or blood products in excess of 500 mL within 84 days of screening
* Lactating females
* Poor or unsuitable venous access
* Treatment with another investigational drug, biological agent, or device within 6 months of screening, or 5 half-lives of the study agent, whichever is longer.
* History of sensitivity to any of the study medications, or metabolite thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation CARDIAC MAGNETIC RESONANCE (CMR) SCANNING
* Orthopnoea of sufficient severity to preclude supine scanning as determined at screening
* Contraindication to magnetic resonance imaging (MRI) contrast agents
* Inability to fit inside scanner due to body size (girth)
* Contraindication for MRI scanning (as assessed by local MRI safety questionnaire), which includes but is not limited to:

  * Intracranial aneurysm clips (except Sugita) or other metallic objects
  * Intra- orbital metal fragments that have not been removed
  * Pacemakers or other implanted cardiac rhythm management/monitoring devices and non-MR conditional heart valves
  * Inner ear implants
  * History of claustrophobia

    99m^TC-PYP OR 99mTC-DPD BONE TRACER RADIOSCINTOGRAPHY
* Orthopnoea of sufficient severity to preclude supine scanning as determined at Screening
* Previous allergic reaction to radioisotope bone tracers
* Previous inclusion in a research protocol involving nuclear medicine, positron emission tomography (PET) or radiological investigations with significant radiation burden (a significant radiation burden being defined as 10 mSv in addition to natural background radiation, in the previous 3 years).

Exclusion Criteria for Group 1

Has any of the following:

* Fulfilment of diagnostic criteria for AL amyloidosis
* TTR polyneuropathy and / or intracranial TTR involvement including ophthalmological disease
* Non-amyloidosis related chronic liver disease (with the exception of Gilbert's syndrome or clinically asymptomatic gallstones)
* Platelet count < 125x10^9 / L

Exclusion criteria for Group 2

* Chronic liver disease or current active liver or biliary disease not attributable to amyloidosis (with the exception of Gilbert's syndrome or asymptomatic gallstones).

Exclusion criteria for Group 3

* Chronic liver disease or current active liver or biliary disease not attributable to amyloidosis (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Platelet count < 75x10^9 /L

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Boston, Massachusetts, United States
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, non-randomized, monthly repeat anti-serum amyloid p component (anti-SAP) treatment study in systemic amyloidosis participants with cardiac dysfunction caused by cardiac amyloidosis.
Pre-assignment Details: Twelve participants were screened; seven were enrolled in to study (six were enrolled in Group 1 and one in Group 2). No participant was enrolled in Group 3. The study was terminated by sponsor due to a change in the benefit:risk profile of GSK2315698+GSK2398852 (anti-SAP treatment).
Groups:
- Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants: Cardiac transthyretin (TTR) amyloidosis (transthyretin amyloid cardiomyopathy [ATTR-CM]) participants with mutant genotypes primarily associated with familial amyloidotic cardiomyopathy (FAC) and wild-type TTR were included. Participants received 6 anti-SAP treatments, consisting of carboxy pyrrolidine hexanoyl pyrrolidine carboxylate (CPHPC) followed by anti-SAP monoclonal antibody (mAb) at monthly intervals. During each anti-SAP treatment, participants received CPHPC intravenous (IV) infusion once daily for up to 72 hours. After 72 hours of CPHPC administration, participants were administered intravenous infusion of anti-SAP mAb over 6-8 hours each on Days 1 and 3. The starting dose level of anti-SAP mAb was 600 milligrams (mg) (divided into 2 infusions of 300 mg). In each treatment session, CPHPC was administered as subcutaneous (SC) injection for 11 days from the day of first dose of anti-SAP mAb.
- Group 2: Post-chemotherapy AL Amyloidosis Participants: Immunoglobin light chain amyloidosis (AL) participants who attained either a very good partial response (VGPR), or complete response (CR), to systemic chemotherapy (including autologous stem cell transplantation) were included. Participants received 6 anti-SAP treatments, consisting of CPHPC followed by anti-SAP mAb at monthly intervals. During each anti-SAP treatment, participants received CPHPC IV infusion once daily for up to 72 hours. After 72 hours of CPHPC administration, participants were administered IV infusion of anti-SAP mAb over 6-8 hours each on Days 1 and 3. The starting dose level of anti-SAP mAb was 600 mg (divided into 2 infusions of 300 mg). In each treatment session, CPHPC was administered by as SC injection for 11 days from the day of first dose of anti-SAP mAb.
- Group 3: Newly Diagnosed Mayo Stage II/IIIa AL Participants: Newly diagnosed Mayo stage II/IIIa AL participants who attained a free light chain CR during the first 3 cycles of first-line chemotherapy where the first cycle was cyclophosphamide, bortezomib, dexamethasone (CyBorD) were planned to be included. Participants were planned to receive 6 anti-SAP treatments, consisting of CPHPC followed by anti-SAP mAb at monthly intervals. During each anti-SAP treatment, participants were planned to receive CPHPC IV infusion once daily for up to 72 hours. After 72 hours of CPHPC administration, participants were planned to administer IV infusion of anti-SAP mAb over 6-8 hours each on Days 1 and 3. The starting dose level of anti-SAP mAb was planned to be 600 mg (divided into 2 infusions of 300 mg). In each treatment session, CPHPC was planned to be administered as SC injection for 11 days from the day of first dose of anti-SAP mAb.
Period: Overall Study
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants | Group 3: Newly Diagnosed Mayo Stage II/IIIa AL Participants
Started | 6 | 1 | 0 (No participant was enrolled in Group-3 due to early termination of the study.)
Completed | 6 | 0 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participant was enrolled in "Group 3: Newly diagnosed Mayo stage II/IIIa AL participant" due to early termination of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants | Group 3: Newly Diagnosed Mayo Stage II/IIIa AL Participants | Total
Number analyzed (Participants) | 6 | 1 | 0 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.3 (3.27) | 67.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants (N=1). |  | 73.3 (4.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 1 | 0 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian/European Heritage | 6 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular (LV) Mass Over Time up to 8-week Follow-up
Description: Left ventricular mass was measured by Cardiac Magnetic Resonance (CMR) imaging to assess reduction in cardiac amyloid load after repeated administration of anti-SAP treatment. Each CMR imaging session took approximately 45-60 minutes, with a maximum scan time inside of the scanner of 90 minutes. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value. Safety Population comprised of all participants who received at least one dose of study treatment (any dose of CPHPC [GSK2315698] or anti-SAP mAb [GSK2398852]).
Time Frame: Baseline (Day -1) and Session 2 Day 24, Session 3 Day 24, Session 4 Day 24, Session 5 Day 24, 8 Weeks Follow-up
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Grams
  Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, Day 24, n=6,0 | 2.505 (19.9174) |
  Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, Day 24, n=6,0 | 4.175 (22.9366) |
  Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, Day 24, n=5,0 | 9.194 (14.4271) |
  Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, Day 24, n=4,0 | 7.955 (19.4341) |
  8 Weeks Follow up, n=6,1 | 0.977 (12.1795) | -32.420 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

2. Primary Outcome: Number of Participants With Any On-treatment Adverse Events (AEs)
Description: AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with any on-treatment AEs are presented.
Time Frame: Up to 56 days after the last dosing session (up to 265 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants | 6 | 1

3. Primary Outcome: Number of Participants With Any Serious Adverse Events (SAEs)
Description: AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, events associated with liver injury and impaired liver function, or any other situation according to medical or scientific judgment were categorized as SAE. Number of participants with any SAEs during study are presented.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants | 2 | 1

4. Primary Outcome: Number of Participants With Abnormal Hematology Values
Description: Blood samples were collected for assessment of hematology parameters, which included platelet count, hemoglobin, hematocrit, erythrocytes, reticulocyte count, Mean corpuscular volume (MCV), Mean corpuscular hemoglobin (MCH), Mean corpuscular hemoglobin concentration (MCHC), neutrophils, lymphocytes, monocytes, eosinophils, leukocytes and basophils. Abnormal laboratory results are categorized as high, low or normal with respect to their normal ranges. Data for worst case post Baseline is presented. Participants having both High and Low values from Normal Ranges at any post-baseline visits for any parameter was counted in both the High and Low categories.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants
  Basophils, high | 2 | 0
  Basophils, normal | 4 | 1
  Basophils, low | 0 | 0
  Eosinophils, high | 3 | 0
  Eosinophils, normal | 3 | 1
  Eosinophils, low | 0 | 0
  Hematocrit, high | 0 | 0
  Hematocrit, normal | 1 | 0
  Hematocrit, low | 5 | 1
  Hemoglobin, high | 0 | 0
  Hemoglobin, normal | 0 | 0
  Hemoglobin, low | 6 | 1
  Lymphocytes, high | 1 | 0
  Lymphocytes, normal | 0 | 0
  Lymphocytes, low | 6 | 1
  MCH, high | 1 | 0
  MCH, normal | 3 | 1
  MCH, low | 3 | 0
  MCHC, high | 3 | 0
  MCHC, normal | 1 | 1
  MCHC, low | 2 | 0
  MCV, high | 1 | 0
  MCV, normal | 4 | 1
  MCV, low | 2 | 0
  Monocytes, high | 2 | 1
  Monocytes, normal | 4 | 0
  Monocytes, low | 0 | 0
  Neutrophils, high | 5 | 1
  Neutrophils, normal | 0 | 0
  Neutrophils, low | 4 | 0
  Platelet count, high | 1 | 0
  Platelet count, normal | 3 | 0
  Platelet count, low | 2 | 1
  Erythrocytes, high | 0 | 0
  Erythrocytes, normal | 0 | 0
  Erythrocytes, low | 6 | 1
  Reticulocytes, high | 1 | 0
  Reticulocytes, normal | 5 | 1
  Reticulocytes, low | 0 | 0
  Leukocytes, high | 2 | 1
  Leukocytes, normal | 3 | 0
  Leukocytes, low | 1 | 0

5. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Values
Description: Blood samples were collected for assessment of clinical chemistry parameters, which included aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), lactate dehydrogenase (LDH), urea, creatinine, glucose, chloride, creatinine kinase, potassium, sodium, calcium, total carbon dioxide (CO2), urate, total and direct bilirubin, total protein and albumin. Abnormal laboratory results are categorized as high, low or normal with respect to their normal ranges. Data for worst case post Baseline is presented. Participants having both High and Low values from Normal Ranges at any post-baseline visits for any parameter was counted in both the High and Low categories.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants
  Glucose, high | 6 | 1
  Glucose, normal | 0 | 0
  Glucose, low | 0 | 0
  Albumin, high | 0 | 0
  Albumin, normal | 2 | 1
  Albumin, low | 4 | 0
  ALP, high | 5 | 0
  ALP, normal | 1 | 1
  ALP, low | 0 | 0
  ALT, high | 2 | 1
  ALT, normal | 4 | 0
  ALT, low | 0 | 0
  AST, high | 4 | 1
  AST, normal | 2 | 0
  AST, low | 0 | 0
  Direct Bilirubin, high | 4 | 1
  Direct Bilirubin, normal | 2 | 0
  Direct Bilirubin, low | 0 | 0
  Total Bilirubin, high | 4 | 0
  Total Bilirubin, normal | 2 | 1
  Total Bilirubin, low | 0 | 0
  Calcium, high | 0 | 0
  Calcium, normal | 4 | 0
  Calcium, low | 2 | 1
  Creatinine Kinase, high | 1 | 0
  Creatinine Kinase, normal | 3 | 1
  Creatinine Kinase, low | 2 | 0
  Chloride, high | 0 | 0
  Chloride, normal | 1 | 0
  Chloride, low | 5 | 1
  CO2, high | 6 | 0
  CO2, normal | 0 | 1
  CO2, low | 4 | 0
  Creatinine, high | 4 | 0
  Creatinine, normal | 2 | 1
  Creatinine, low | 0 | 0
  Potassium, high | 2 | 0
  Potassium, normal | 3 | 1
  Potassium, low | 2 | 0
  LDH, high | 6 | 1
  LDH, normal | 0 | 0
  LDH, low | 0 | 0
  Protein, high | 0 | 0
  Protein, normal | 0 | 0
  Protein, low | 6 | 1
  Sodium, high | 1 | 0
  Sodium, normal | 5 | 1
  Sodium, low | 0 | 0
  Urate, high | 5 | 1
  Urate, normal | 1 | 0
  Urate, low | 0 | 0
  Urea, high | 6 | 1
  Urea, normal | 0 | 0
  Urea, low | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Urinalysis Results
Description: Urine samples were collected to assess potential of hydrogen (pH), specific gravity, albumin excretion rate, creatinine excretion rate and protein excretion rate. Abnormal urinalysis results are categorized as high, low or normal with respect to their normal ranges. Data for worst case post Baseline is presented. Participants having both High and Low values from Normal Ranges at any post-baseline visits for any parameter was counted in both the High and Low categories.
Time Frame: Up to the end of study (Up to 369 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants
  pH, high, n=6,1 | 0 | 0
  pH, normal, n=6,1 | 6 | 1
  pH, low, n=6,1 | 0 | 0
  Specific gravity, high, n=1,0: number analyzed (Participants) | 1 | 0
  Specific gravity, high, n=1,0 | 0 |
  Specific gravity, normal, n=1,0: number analyzed (Participants) | 1 | 0
  Specific gravity, normal, n=1,0 | 1 |
  Specific gravity, low, n=1,0: number analyzed (Participants) | 1 | 0
  Specific gravity, low, n=1,0 | 0 |
  Albumin excretion rate, high, n=6,1 | 0 | 0
  Albumin excretion rate, normal, n=6,1 | 6 | 1
  Albumin excretion rate, low, n=6,1 | 0 | 0
  Creatinine excretion rate, high, n=6,1 | 1 | 0
  Creatinine excretion rate, normal, n=6,1 | 1 | 1
  Creatinine excretion rate, low, n=6,1 | 5 | 0
  Protein excretion rate, high, n=6,1 | 4 | 1
  Protein excretion rate, normal, n=6,1 | 2 | 0
  Protein excretion rate, low, n=6,1 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Urinalysis Results for Character Parameters
Description: Urine samples were collected to assess character parameters which included Cellular Casts, Erythrocytes, Glucose, Ketones, Leukocytes and Occult Blood. Number of participants with abnormal urinalysis results are presented. Data for worst case post Baseline is presented.
Time Frame: Up to the end of study (Up to 369 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants
  Cellular casts, n=5,1: number analyzed (Participants) | 5 | 1
  Cellular casts, n=5,1 | 0 | 0
  Erythrocytes , n=6,1 | 6 | 1
  Glucose, n=6,1 | 1 | 0
  Ketones, n=6,1 | 0 | 0
  Leukocytes, n=6,1 | 6 | 1
  Occult blood, n=6,1 | 2 | 1

8. Primary Outcome: Number of Participants With Body Temperature Shifts From Baseline Relative to Potential Clinical Importance (PCI) Criteria
Description: Vital signs including body temperature was measured after participants rested in semi-supine position for at least 5 minutes. Number of participants with shifts in body temperature from Baseline to worst case post Baseline relative to PCI criteria have been presented. PCI results were categorized as to high, to low and to normal/no change with reference to PCI criteria. PCI criteria for body temperature was: high: >37.5 degree Celsius; low: not applicable.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants
  To high | 2 | 0
  To normal/No change | 4 | 1
  To low | 0 | 0

9. Primary Outcome: Number of Participants With Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Shifts From Baseline Relative to PCI Criteria
Description: Vital signs including SBP and DBP were measured after participants rested in semi-supine position for at least 5 minutes. Number of participants with shifts in SBP and DBP from baseline to worst case post baseline relative to PCI criteria have been presented. PCI results were categorized as to high, to low and to normal/no change with reference to PCI criteria. PCI criteria for SBP was: high: >180 millimeter of mercury (mmHg); low: <90 mmHg. PCI criteria for DBP was: high: >110 mmHg; low: <30 mmHg.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants
  SBP, To high | 0 | 0
  SBP, To normal/No change | 1 | 1
  SBP, To low | 5 | 0
  DBP, To high | 0 | 0
  DBP, To normal/No change | 6 | 1
  DBP, To low | 0 | 0

10. Primary Outcome: Number of Participants With Pulse Rate Shifts From Baseline Relative to PCI Criteria
Description: Vital signs including pulse rate were measured after participants rested in semi-supine position for at least 5 minutes. Number of participants with shifts in pulse rate from baseline to worst case post baseline relative to PCI criteria have been presented. PCI results were categorized as to high, to low and to normal/no change with reference to its PCI criteria. PCI criteria for pulse rate was: high: >140 beats per minute (bpm); low: <35 bpm.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants
  To high | 0 | 0
  To normal/No change | 6 | 1
  To low | 0 | 0

11. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve-lead ECGs were performed during the study using an automated ECG machine. The number of participants with worst case post-Baseline abnormal ECG findings were reported and categorized as abnormal-clinically significant and abnormal-not clinically significant.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants
  Abnormal-Clinically significant | 0 | 0
  Abnormal-Not Clinically significant | 6 | 1

12. Primary Outcome: Number of Participants With Abnormalities During Cardiac Monitoring
Description: Lead II telemetry and cardiac monitoring devices were used for electrical cardiac monitoring during the study. The number of participants with worst case post-Baseline abnormalities during cardiac monitoring as per investigator's assessment have been reported and categorized as Abnormal-clinically significant and Abnormal-not clinically significant.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population. Only those participants with data available at the specified time point was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 5 | 1
Participants
  Abnormal-Clinically significant | 2 | 0
  Abnormal-Not Clinically significant | 3 | 1

13. Primary Outcome: Number of Participants for Which Unscheduled Echocardiography (ECHO) Was Performed for Safety Reasons
Description: Echocardiography was performed by a qualified echocardiographer or cardiologist during the study. Number of participants with unscheduled echocardiograms performed for safety reasons have been presented.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population. Only those participants with data available at the specified time point was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 2 | 0
Participants | 2 |

14. Primary Outcome: Number of Participants With Skin Rashes
Description: Skin rash was an event of special interest. Only Rashes that were associated with study drug were categorised as Rash for Common Terminology Criteria for Adverse Events (CTCAE) and are presented. Number of participants with on-treatment skin rash AEs are presented.
Time Frame: Up to 56 days after the last dosing session (up to 265 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants | 4 | 0

15. Primary Outcome: Number of Participants With Skin Rashes Classified Using CTCAE
Description: Skin rash was an event of special interest. All the events of rashes were graded for their severity using CTCAE version 4.0 . Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life threatening, Grade 5: death. Higher the grade, more severe the symptoms. Only Rashes that were associated with study drug were categorised as Rash for CTCAE and are presented here. Number of participants with skin rashes classified by their maximum grade are presented.
Time Frame: Up to 56 days after the last dosing session (up to 265 days)
Population: Safety Population. Only those participants with data available at the specified time point was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 4 | 0
Participants
  Grade 1 | 3 |
  Grade 2 | 1 |
  Grade 3 | 0 |
  Grade 4 | 0 |
  Grade 5 | 0 |

16. Secondary Outcome: Number of Participants With Abnormalities in Histopathological Examination of Skin Biopsies
Description: Skin biopsy samples were collected for histopathological examination only on any rash development (>= Grade 1) as decided by clinical judgment of the Investigator and/or dermatologist. Number of participants with abnormalities in histopathological examination of skin biopsies are presented.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants | 2 | 0

17. Secondary Outcome: Number of Participants With Abnormalities in Immunohistochemical Examination of Skin Biopsies
Description: Skin biopsy samples were collected for immunohistochemical examination only on any rash development (>= Grade 1) as decided by clinical judgment of the Investigator and/or dermatologist. Number of participants with abnormalities in immunohistochemical examination of skin biopsies are presented.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Participants | 2 | 0

18. Secondary Outcome: Number of Participants With Abnormalities in Histopathological Examination of Blood Biomarkers
Description: Blood samples were to be collected along with each skin biopsy sample for histopathological examination of blood biomarkers only on any rash development (>= Grade 1) as decided by clinical judgment of the Investigator and/or dermatologist.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population. Data was not collected due to project termination.
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Number of Participants With Abnormalities in Immunohistochemical Examination of Blood Biomarkers
Description: Blood samples were to be collected along with each skin biopsy sample for immunohistochemical examination of blood biomarkers only on any rash development (>= Grade 1) as decided by clinical judgment of the Investigator and/or dermatologist.
Time Frame: Up to the end of study (Up to 369 days)
Population: Safety Population. Data was not collected due to project termination.
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in Plasma Cytokines Over Time
Description: Blood samples were collected for assessment of plasma cytokines biomarkers which included Tumor Necrosis Factor (TNF), Interleukin 1 beta (IL-1 beta), IL-6, IL-10, Interferon gamma (INF gamma), IL-12, IL-13, IL-2, IL-4 and IL-8. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value. Absolute values below the lower limit of quantification (LLQ) were imputed with half the LLQ and those above the upper limit of quantification (ULQ) were imputed with the ULQ.
Time Frame: Baseline (Day -1) and Session 1: Day 1 (predose, 1,3,6 hours), Day 2, Day 3 (predose, 1,3,6 hours), Day 4, Day 5; Session 2 to 6: Day -2, Day 1 (predose, 1,3,6 hours), Day 2, Day 3 (predose, 1,3,6 hours), Day 4, Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nanograms per liter (ng/L)
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Nanograms per liter (ng/L)
  IL-1 beta, Session 1, Day 1, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-1 beta, Session 1, Day 1, 1 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-1 beta, Session 1, Day 1, 3 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-1 beta, Session 1, Day 1, 6 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-1 beta, Session 1, Day 2, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-1 beta, Session 1, Day 3, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-1 beta, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 1, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 1, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 1, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 1, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 1, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day -2, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 2, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 3, predose, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 2, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 3, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 3, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 3, predose, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 3, 1 hour, n=6,0 | 0.293 (0.7185) |
  IL-1 beta, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-1 beta, Session 3, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 1, predose, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 1, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 1, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 1, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 3, predose, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 3, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 3, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 3, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-1 beta, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  IL-1 beta, Session 4, Day 4, n=5,0 | 0.504 (1.1270) |
  IL-1 beta, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 4, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 3, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 4, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 5, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 3, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 4, n=4,0 | 0.000 (0.0000) |
  IL-1 beta, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-1 beta, Session 6, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-6, Session 1, Day 1, predose, n=6,1 | 0.275 (0.4711) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-6, Session 1, Day 1, 1 hour, n=6,1 | -0.080 (0.7723) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-6, Session 1, Day 1, 3 hour, n=6,1 | -0.727 (1.2035) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-6, Session 1, Day 1, 6 hour, n=6,1 | -1.077 (1.2511) | 2.880 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-6, Session 1, Day 2, n=6,1 | 6.278 (6.3567) | 29.030 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-6, Session 1, Day 3, predose, n=6,1 | 7.688 (8.8639) | 16.980 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-6, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 1, Day 3, 1 hour, n=6,0 | 6.857 (10.5934) |
  IL-6, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 1, Day 3, 3 hour, n=6,0 | 0.827 (3.5790) |
  IL-6, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 1, Day 3, 6 hour, n=6,0 | 0.932 (5.5637) |
  IL-6, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 1, Day 4, n=6,0 | 5.453 (3.6039) |
  IL-6, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 1, Day 5, n=6,0 | 3.245 (3.3934) |
  IL-6, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day -2, n=6,0 | 0.393 (0.5250) |
  IL-6, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 1, predose, n=6,0 | 0.632 (1.2026) |
  IL-6, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 1, 1 hour, n=6,0 | 0.025 (0.7117) |
  IL-6, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 1, 3 hour, n=6,0 | -0.860 (1.0909) |
  IL-6, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 1, 6 hour, n=6,0 | -0.282 (1.7148) |
  IL-6, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 2, n=6,0 | 21.590 (27.1214) |
  IL-6, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 3, predose, n=6,0 | 11.365 (11.4140) |
  IL-6, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 3, 1 hour, n=6,0 | 7.517 (8.6084) |
  IL-6, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 3, 3 hour, n=6,0 | 3.460 (5.0176) |
  IL-6, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 3, 6 hour, n=6,0 | 0.723 (4.5392) |
  IL-6, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 4, n=6,0 | 4.580 (5.9326) |
  IL-6, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 2, Day 5, n=6,0 | 6.395 (5.2800) |
  IL-6, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 3, Day -2, n=5,0 | 0.148 (0.8211) |
  IL-6, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 1, predose, n=6,0 | 0.782 (1.5023) |
  IL-6, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 1, 1 hour, n=6,0 | 0.268 (1.4865) |
  IL-6, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 1, 3 hour, n=6,0 | 0.062 (2.5899) |
  IL-6, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 1, 6 hour, n=6,0 | -0.918 (1.2591) |
  IL-6, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 3, Day 2, n=5,0 | 17.608 (29.2558) |
  IL-6, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 3, predose, n=6,0 | 11.872 (8.7413) |
  IL-6, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 3, 1 hour, n=6,0 | 5.835 (3.8271) |
  IL-6, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 3, 3 hour, n=6,0 | 1.742 (1.9174) |
  IL-6, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 3, 6 hour, n=6,0 | 0.063 (2.2072) |
  IL-6, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 4, n=6,0 | 4.667 (6.9875) |
  IL-6, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-6, Session 3, Day 5, n=6,0 | 5.570 (2.6004) |
  IL-6, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day -2, n=5,0 | 0.892 (0.8423) |
  IL-6, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 1, predose, n=5,0 | 1.486 (0.8702) |
  IL-6, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 1, 1 hour, n=5,0 | 0.926 (0.7103) |
  IL-6, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 1, 3 hour, n=5,0 | -0.026 (0.1599) |
  IL-6, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 1, 6 hour, n=5,0 | -1.028 (1.3685) |
  IL-6, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 2, n=5,0 | 5.720 (11.3851) |
  IL-6, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 3, predose, n=5,0 | 10.924 (6.5370) |
  IL-6, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 3, 1 hour, n=5,0 | 4.486 (2.0420) |
  IL-6, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 3, 3 hour, n=5,0 | 1.446 (1.5368) |
  IL-6, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 3, 6 hour, n=5,0 | -0.116 (1.7948) |
  IL-6, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  IL-6, Session 4, Day 4, n=5,0 | 5.756 (6.8645) |
  IL-6, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 4, Day 5, n=4,0 | 4.388 (3.7765) |
  IL-6, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day -2, n=4,0 | 0.027 (0.8164) |
  IL-6, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 1, predose, n=4,0 | 0.865 (0.9927) |
  IL-6, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 1, 1 hour, n=4,0 | -0.007 (1.3219) |
  IL-6, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 1, 3 hour, n=4,0 | -0.423 (1.5816) |
  IL-6, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 1, 6 hour, n=4,0 | -1.213 (1.5189) |
  IL-6, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 2, n=4,0 | 0.905 (4.0920) |
  IL-6, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 3, predose, n=4,0 | 7.323 (4.8265) |
  IL-6, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 3, 1 hour, n=4,0 | 4.240 (3.6214) |
  IL-6, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 3, 3 hour, n=4,0 | -0.125 (0.7543) |
  IL-6, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 3, 6 hour, n=4,0 | -1.390 (1.3301) |
  IL-6, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 4, n=4,0 | 3.598 (5.7476) |
  IL-6, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 5, Day 5, n=4,0 | 6.533 (2.6812) |
  IL-6, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day -2, n=4,0 | 1.383 (1.8535) |
  IL-6, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 1, predose, n=4,0 | 0.565 (1.4007) |
  IL-6, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 1, 1 hour, n=4,0 | 0.077 (1.1200) |
  IL-6, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 1, 3 hour, n=4,0 | -0.413 (1.4416) |
  IL-6, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 1, 6 hour, n=4,0 | -1.165 (0.9786) |
  IL-6, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 2, n=4,0 | 0.932 (4.0340) |
  IL-6, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 3, predose, n=4,0 | 15.008 (13.0010) |
  IL-6, Session 6, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 3, 1 hour, n=4,0 | 10.083 (9.2076) |
  IL-6, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 3, 3 hour, n=4,0 | 1.435 (1.7505) |
  IL-6, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 3, 6 hour, n=4,0 | -1.005 (1.3522) |
  IL-6, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 4, n=4,0 | 1.740 (3.2649) |
  IL-6, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-6, Session 6, Day 5, n=4,0 | 7.190 (3.8811) |
  IL-10, Session 1, Day 1, predose, n=6,1 | -0.067 (0.1633) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-10, Session 1, Day 1, 1 hour, n=6,1 | 0.105 (0.1663) | 8.580 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-10, Session 1, Day 1, 3 hour, n=6,1 | 0.763 (0.4804) | 5.260 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-10, Session 1, Day 1, 6 hour, n=6,1 | 1.710 (1.4719) | 6.020 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-10, Session 1, Day 2, n=6,1 | -0.005 (0.2436) | 1.150 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-10, Session 1, Day 3, predose, n=6,1 | 0.040 (0.3347) | 1.280 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-10, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 1, Day 3, 1 hour, n=6,0 | 0.670 (1.0153) |
  IL-10, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 1, Day 3, 3 hour, n=6,0 | 0.065 (0.3896) |
  IL-10, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 1, Day 3, 6 hour, n=6,0 | 0.002 (0.0041) |
  IL-10, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 1, Day 4, n=6,0 | -0.067 (0.1633) |
  IL-10, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 1, Day 5, n=6,0 | -0.067 (0.1633) |
  IL-10, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day -2, n=6,0 | -0.067 (0.1633) |
  IL-10, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 1, predose, n=6,0 | 0.002 (0.0041) |
  IL-10, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 1, 1 hour, n=6,0 | 0.612 (0.8293) |
  IL-10, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 1, 3 hour, n=6,0 | 1.132 (1.1748) |
  IL-10, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 1, 6 hour, n=6,0 | 0.785 (0.5189) |
  IL-10, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 2, n=6,0 | 0.012 (0.2757) |
  IL-10, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 3, predose, n=6,0 | 0.233 (0.5618) |
  IL-10, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 3, 1 hour, n=6,0 | 0.775 (1.1274) |
  IL-10, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 3, 3 hour, n=6,0 | 0.782 (0.8451) |
  IL-10, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 3, 6 hour, n=6,0 | 0.015 (0.0367) |
  IL-10, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 4, n=6,0 | -0.005 (0.0122) |
  IL-10, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 2, Day 5, n=6,0 | 0.110 (0.2122) |
  IL-10, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 3, Day -2, n=5,0 | 0.032 (0.3422) |
  IL-10, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 1, predose, n=6,0 | -0.067 (0.1633) |
  IL-10, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 1, 1 hour, n=6,0 | 0.228 (0.2328) |
  IL-10, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 1, 3 hour, n=6,0 | 1.185 (1.1559) |
  IL-10, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 1, 6 hour, n=6,0 | 0.495 (0.6641) |
  IL-10, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 3, Day 2, n=5,0 | -0.080 (0.1789) |
  IL-10, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 3, predose, n=6,0 | -0.067 (0.1633) |
  IL-10, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 3, 1 hour, n=6,0 | 0.450 (0.6048) |
  IL-10, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 3, 3 hour, n=6,0 | 0.322 (0.5322) |
  IL-10, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 3, 6 hour, n=6,0 | 0.092 (0.1542) |
  IL-10, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 4, n=6,0 | -0.067 (0.1633) |
  IL-10, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-10, Session 3, Day 5, n=6,0 | -0.067 (0.1633) |
  IL-10, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day -2, n=5,0 | -0.080 (0.1789) |
  IL-10, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 1, predose, n=5,0 | -0.080 (0.1789) |
  IL-10, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 1, 1 hour, n=5,0 | 0.758 (1.4466) |
  IL-10, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 1, 3 hour, n=5,0 | 3.868 (6.3123) |
  IL-10, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 1, 6 hour, n=5,0 | 0.868 (0.9281) |
  IL-10, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 2, n=5,0 | -0.080 (0.1789) |
  IL-10, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 3, predose, n=5,0 | 0.022 (0.0492) |
  IL-10, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 3, 1 hour, n=5,0 | 0.808 (1.0592) |
  IL-10, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 3, 3 hour, n=5,0 | 0.598 (0.6549) |
  IL-10, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 3, 6 hour, n=5,0 | 0.184 (0.4284) |
  IL-10, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  IL-10, Session 4, Day 4, n=5,0 | -0.080 (0.1789) |
  IL-10, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 4, Day 5, n=4,0 | -0.100 (0.2000) |
  IL-10, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day -2, n=4,0 | -0.100 (0.2000) |
  IL-10, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 1, predose, n=4,0 | -0.100 (0.2000) |
  IL-10, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 1, 1 hour, n=4,0 | 2.485 (4.8507) |
  IL-10, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 1, 3 hour, n=4,0 | 3.828 (6.5828) |
  IL-10, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 1, 6 hour, n=4,0 | 1.120 (1.5607) |
  IL-10, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 2, n=4,0 | -0.100 (0.2000) |
  IL-10, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 3, predose, n=4,0 | 0.393 (0.4774) |
  IL-10, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 3, 1 hour, n=4,0 | 0.950 (0.9330) |
  IL-10, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 3, 3 hour, n=4,0 | 1.060 (0.9783) |
  IL-10, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 3, 6 hour, n=4,0 | 0.663 (0.6663) |
  IL-10, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 4, n=4,0 | 0.210 (0.4267) |
  IL-10, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 5, Day 5, n=4,0 | 0.025 (0.0500) |
  IL-10, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day -2, n=4,0 | -0.100 (0.2000) |
  IL-10, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 1, predose, n=4,0 | -0.100 (0.2000) |
  IL-10, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 1, 1 hour, n=4,0 | 0.333 (0.9506) |
  IL-10, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 1, 3 hour, n=4,0 | 1.738 (2.5365) |
  IL-10, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 1, 6 hour, n=4,0 | 1.418 (1.7245) |
  IL-10, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 2, n=4,0 | -0.100 (0.2000) |
  IL-10, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 3, predose, n=4,0 | 0.015 (0.0300) |
  IL-10, Session 6, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 3, 1 hour, n=4,0 | 0.753 (1.4004) |
  IL-10, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 3, 3 hour, n=4,0 | 0.675 (1.1466) |
  IL-10, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 3, 6 hour, n=4,0 | 0.220 (0.2723) |
  IL-10, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 4, n=4,0 | -0.100 (0.2000) |
  IL-10, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-10, Session 6, Day 5, n=4,0 | 0.023 (0.0450) |
  TNF, Session 1, Day 1, predose, n=6,1 | 0.055 (0.4378) | 0.320 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  TNF, Session 1, Day 1, 1 hour, n=6,1 | 0.007 (0.7159) | 0.100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  TNF, Session 1, Day 1, 3 hour, n=6,1 | -0.180 (0.7430) | 0.880 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  TNF, Session 1, Day 1, 6 hour, n=6,1 | -0.132 (0.8145) | 2.300 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  TNF, Session 1, Day 2, n=6,1 | 1.920 (1.5379) | 5.130 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  TNF, Session 1, Day 3, predose, n=6,1 | 1.453 (1.3405) | 3.010 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  TNF, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 1, Day 3, 1 hour, n=6,0 | 1.240 (0.9968) |
  TNF, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 1, Day 3, 3 hour, n=6,0 | 0.797 (1.0229) |
  TNF, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 1, Day 3, 6 hour, n=6,0 | 0.460 (0.9373) |
  TNF, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 1, Day 4, n=6,0 | 1.088 (1.2874) |
  TNF, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 1, Day 5, n=6,0 | 1.577 (1.5915) |
  TNF, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day -2, n=6,0 | 0.167 (0.9735) |
  TNF, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 1, predose, n=6,0 | 0.233 (0.8351) |
  TNF, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 1, 1 hour, n=6,0 | 0.133 (1.0259) |
  TNF, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 1, 3 hour, n=6,0 | 0.015 (1.0940) |
  TNF, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 1, 6 hour, n=6,0 | -0.100 (1.2625) |
  TNF, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 2, n=6,0 | 1.523 (1.6646) |
  TNF, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 3, predose, n=6,0 | 2.143 (1.5642) |
  TNF, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 3, 1 hour, n=6,0 | 1.682 (1.3855) |
  TNF, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 3, 3 hour, n=6,0 | 1.133 (0.9970) |
  TNF, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 3, 6 hour, n=6,0 | 0.503 (1.0718) |
  TNF, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 4, n=6,0 | 1.397 (2.1712) |
  TNF, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 2, Day 5, n=6,0 | 1.968 (1.4560) |
  TNF, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 3, Day -2, n=5,0 | 0.098 (1.2163) |
  TNF, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 1, predose, n=6,0 | 0.497 (0.9650) |
  TNF, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 1, 1 hour, n=6,0 | -0.297 (0.9572) |
  TNF, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 1, 3 hour, n=6,0 | -0.198 (0.9246) |
  TNF, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 1, 6 hour, n=6,0 | -0.167 (1.2317) |
  TNF, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 3, Day 2, n=5,0 | 0.446 (1.1212) |
  TNF, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 3, predose, n=6,0 | 1.267 (1.1583) |
  TNF, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 3, 1 hour, n=6,0 | 0.513 (1.1234) |
  TNF, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 3, 3 hour, n=6,0 | 0.128 (1.0706) |
  TNF, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 3, 6 hour, n=6,0 | 0.233 (1.2605) |
  TNF, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 4, n=6,0 | 0.585 (1.6017) |
  TNF, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  TNF, Session 3, Day 5, n=6,0 | 0.997 (1.3819) |
  TNF, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day -2, n=5,0 | -0.208 (0.5949) |
  TNF, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 1, predose, n=5,0 | -0.214 (0.8527) |
  TNF, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 1, 1 hour, n=5,0 | 0.160 (1.5494) |
  TNF, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 1, 3 hour, n=5,0 | 0.218 (1.5011) |
  TNF, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 1, 6 hour, n=5,0 | -0.412 (1.1373) |
  TNF, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 2, n=5,0 | -0.122 (0.6977) |
  TNF, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 3, predose, n=5,0 | 0.606 (0.5265) |
  TNF, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 3, 1 hour, n=5,0 | 0.100 (0.5074) |
  TNF, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 3, 3 hour, n=5,0 | 0.098 (0.7172) |
  TNF, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 3, 6 hour, n=5,0 | -0.702 (0.5368) |
  TNF, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  TNF, Session 4, Day 4, n=5,0 | -0.270 (0.7576) |
  TNF, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 4, Day 5, n=4,0 | 0.095 (0.4456) |
  TNF, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day -2, n=4,0 | -0.350 (0.5814) |
  TNF, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 1, predose, n=4,0 | -0.320 (0.6703) |
  TNF, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 1, 1 hour, n=4,0 | -0.130 (1.2227) |
  TNF, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 1, 3 hour, n=4,0 | -0.055 (1.0728) |
  TNF, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 1, 6 hour, n=4,0 | -0.513 (1.1003) |
  TNF, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 2, n=4,0 | -0.498 (0.9752) |
  TNF, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 3, predose, n=4,0 | 0.147 (0.8951) |
  TNF, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 3, 1 hour, n=4,0 | -0.188 (0.7406) |
  TNF, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 3, 3 hour, n=4,0 | -0.378 (0.9306) |
  TNF, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 3, 6 hour, n=4,0 | -0.630 (0.7857) |
  TNF, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 4, n=4,0 | -0.100 (1.0725) |
  TNF, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 5, Day 5, n=4,0 | 0.168 (0.3909) |
  TNF, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day -2, n=4,0 | -0.428 (1.3664) |
  TNF, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 1, predose, n=4,0 | -0.238 (1.3158) |
  TNF, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 1, 1 hour, n=4,0 | -0.303 (1.3853) |
  TNF, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 1, 3 hour, n=4,0 | -0.145 (1.8684) |
  TNF, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 1, 6 hour, n=4,0 | -0.500 (1.4020) |
  TNF, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 2, n=4,0 | -0.000 (1.3253) |
  TNF, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 3, predose, n=4,0 | 0.278 (1.9987) |
  TNF, Session 6, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 3, 1 hour, n=4,0 | -0.195 (1.6007) |
  TNF, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 3, 3 hour, n=4,0 | -0.385 (1.4669) |
  TNF, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 3, 6 hour, n=4,0 | -0.585 (1.3026) |
  TNF, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 4, n=4,0 | -0.368 (1.1280) |
  TNF, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  TNF, Session 6, Day 5, n=4,0 | 0.322 (1.2795) |
  INF gamma, Session 1, Day 1, predose, n=6,1 | 0.075 (1.6224) | 1.860 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  INF gamma, Session 1, Day 1, 1 hour, n=6,1 | -1.373 (2.1255) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  INF gamma, Session 1, Day 1, 3 hour, n=6,1 | -3.298 (3.1409) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  INF gamma, Session 1, Day 1, 6 hour, n=6,1 | -3.298 (3.1409) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  INF gamma, Session 1, Day 2, n=6,1 | 1.713 (7.5955) | 1.930 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  INF gamma, Session 1, Day 3, predose, n=6,1 | 17.122 (27.3980) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  INF gamma, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 1, Day 3, 1 hour, n=6,0 | 12.118 (22.0807) |
  INF gamma, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 1, Day 3, 3 hour, n=6,0 | 7.150 (18.4949) |
  INF gamma, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 1, Day 3, 6 hour, n=6,0 | 0.538 (8.5114) |
  INF gamma, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 1, Day 4, n=6,0 | 3.242 (12.2847) |
  INF gamma, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 1, Day 5, n=6,0 | 19.502 (38.3215) |
  INF gamma, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day -2, n=6,0 | -1.045 (3.4175) |
  INF gamma, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 1, predose, n=6,0 | 0.452 (3.5018) |
  INF gamma, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 1, 1 hour, n=6,0 | 0.145 (3.2180) |
  INF gamma, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 1, 3 hour, n=6,0 | -1.833 (1.3991) |
  INF gamma, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 1, 6 hour, n=6,0 | -3.072 (2.6378) |
  INF gamma, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 2, n=6,0 | -2.660 (3.5043) |
  INF gamma, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 3, predose, n=6,0 | -1.045 (2.2260) |
  INF gamma, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 3, 1 hour, n=6,0 | -1.580 (2.5672) |
  INF gamma, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 3, 3 hour, n=6,0 | -2.473 (2.5631) |
  INF gamma, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 3, 6 hour, n=6,0 | -3.298 (3.1409) |
  INF gamma, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 4, n=6,0 | -2.572 (3.4040) |
  INF gamma, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 2, Day 5, n=6,0 | -1.993 (2.8977) |
  INF gamma, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 3, Day -2, n=5,0 | -2.190 (3.9839) |
  INF gamma, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 1, predose, n=6,0 | -1.035 (4.4739) |
  INF gamma, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 1, 1 hour, n=6,0 | -2.180 (3.8365) |
  INF gamma, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 1, 3 hour, n=6,0 | -3.298 (3.1409) |
  INF gamma, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 1, 6 hour, n=6,0 | -3.298 (3.1409) |
  INF gamma, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 3, Day 2, n=5,0 | -2.936 (3.7855) |
  INF gamma, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 3, predose, n=6,0 | -2.948 (2.3737) |
  INF gamma, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 3, 1 hour, n=6,0 | -3.298 (3.1409) |
  INF gamma, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 3, 3 hour, n=6,0 | -3.298 (3.1409) |
  INF gamma, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 3, 6 hour, n=6,0 | -3.298 (3.1409) |
  INF gamma, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 4, n=6,0 | -3.048 (3.1886) |
  INF gamma, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  INF gamma, Session 3, Day 5, n=6,0 | -2.752 (3.2989) |
  INF gamma, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day -2, n=5,0 | 0.298 (5.3631) |
  INF gamma, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 1, predose, n=5,0 | -0.760 (4.2290) |
  INF gamma, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 1, 1 hour, n=5,0 | -1.240 (4.3736) |
  INF gamma, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 1, 3 hour, n=5,0 | -2.778 (3.9570) |
  INF gamma, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 1, 6 hour, n=5,0 | -3.274 (3.5110) |
  INF gamma, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 2, n=5,0 | -3.274 (3.5110) |
  INF gamma, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 3, predose, n=5,0 | -2.836 (2.6051) |
  INF gamma, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 3, 1 hour, n=5,0 | -3.274 (3.5110) |
  INF gamma, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 3, 3 hour, n=5,0 | -3.274 (3.5110) |
  INF gamma, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 3, 6 hour, n=5,0 | -3.274 (3.5110) |
  INF gamma, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  INF gamma, Session 4, Day 4, n=5,0 | -3.274 (3.5110) |
  INF gamma, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 4, Day 5, n=4,0 | -2.910 (3.1667) |
  INF gamma, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day -2, n=4,0 | -0.930 (3.5480) |
  INF gamma, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 1, predose, n=4,0 | -1.328 (2.1878) |
  INF gamma, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 1, 1 hour, n=4,0 | -1.423 (1.9828) |
  INF gamma, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 1, 3 hour, n=4,0 | -2.725 (2.8230) |
  INF gamma, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 1, 6 hour, n=4,0 | -3.373 (4.0462) |
  INF gamma, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 2, n=4,0 | -3.373 (4.0462) |
  INF gamma, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 3, predose, n=4,0 | 0.753 (4.9155) |
  INF gamma, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 3, 1 hour, n=4,0 | 0.203 (4.5195) |
  INF gamma, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 3, 3 hour, n=4,0 | -1.388 (4.8505) |
  INF gamma, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 3, 6 hour, n=4,0 | -2.838 (4.4804) |
  INF gamma, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 4, n=4,0 | -1.653 (6.0355) |
  INF gamma, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 5, Day 5, n=4,0 | -0.615 (2.9091) |
  INF gamma, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day -2, n=4,0 | -2.625 (4.4662) |
  INF gamma, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 1, predose, n=4,0 | -2.668 (4.4299) |
  INF gamma, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 1, 1 hour, n=4,0 | -2.823 (4.3091) |
  INF gamma, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 1, 3 hour, n=4,0 | -3.373 (4.0462) |
  INF gamma, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 1, 6 hour, n=4,0 | -3.373 (4.0462) |
  INF gamma, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 2, n=4,0 | -3.373 (4.0462) |
  INF gamma, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 3, predose, n=4,0 | -1.988 (5.0857) |
  INF gamma, Session 6, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 3, 1 hour, n=4,0 | -3.018 (4.1848) |
  INF gamma, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 3, 3 hour, n=4,0 | -3.373 (4.0462) |
  INF gamma, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 3, 6 hour, n=4,0 | -3.373 (4.0462) |
  INF gamma, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 4, n=4,0 | -3.373 (4.0462) |
  INF gamma, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  INF gamma, Session 6, Day 5, n=4,0 | -3.373 (4.0462) |
  IL-12, Session 1, Day 1, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-12, Session 1, Day 1, 1 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-12, Session 1, Day 1, 3 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-12, Session 1, Day 1, 6 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-12, Session 1, Day 2, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-12, Session 1, Day 3, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-12, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 1, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 1, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 1, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 1, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 1, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day -2, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 2, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 3, predose, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 2, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 3, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 3, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 3, predose, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-12, Session 3, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 1, predose, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 1, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 1, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 1, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 3, predose, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 3, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 3, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 3, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  IL-12, Session 4, Day 4, n=5,0 | 0.000 (0.0000) |
  IL-12, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 4, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 3, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 4, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 5, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 3, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 4, n=4,0 | 0.000 (0.0000) |
  IL-12, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-12, Session 6, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 1, Day 1, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-13, Session 1, Day 1, 1 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-13, Session 1, Day 1, 3 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-13, Session 1, Day 1, 6 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-13, Session 1, Day 2, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-13, Session 1, Day 3, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-13, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 1, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 1, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 1, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 1, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 1, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day -2, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 2, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 3, predose, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 2, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 3, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 3, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 3, predose, n=6,0 | 0.333 (0.8165) |
  IL-13, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-13, Session 3, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 1, predose, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 1, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 1, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 1, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 3, predose, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 3, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 3, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 3, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  IL-13, Session 4, Day 4, n=5,0 | 0.000 (0.0000) |
  IL-13, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 4, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 3, 1 hour, n=4,0 | 0.283 (0.5650) |
  IL-13, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 4, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 5, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-13, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 4, n=4,0 | 0.488 (0.9750) |
  IL-13, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-13, Session 6, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 1, Day 1, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-2, Session 1, Day 1, 1 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-2, Session 1, Day 1, 3 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-2, Session 1, Day 1, 6 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-2, Session 1, Day 2, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-2, Session 1, Day 3, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-2, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 1, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 1, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 1, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 1, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 1, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day -2, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 2, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 3, predose, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 2, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 3, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 3, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 3, predose, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-2, Session 3, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 1, predose, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 1, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 1, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 1, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 3, predose, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 3, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 3, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 3, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  IL-2, Session 4, Day 4, n=5,0 | 0.000 (0.0000) |
  IL-2, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 4, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 3, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 4, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 5, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 3, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 4, n=4,0 | 0.000 (0.0000) |
  IL-2, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-2, Session 6, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 1, Day 1, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-4, Session 1, Day 1, 1 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-4, Session 1, Day 1, 3 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-4, Session 1, Day 1, 6 hour, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-4, Session 1, Day 2, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-4, Session 1, Day 3, predose, n=6,1 | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-4, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 1, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 1, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 1, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 1, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 1, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day -2, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 2, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 3, predose, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 2, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 3, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 1, predose, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 1, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 1, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 1, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 3, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 3, predose, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 3, 1 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 3, 3 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 3, 6 hour, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 4, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-4, Session 3, Day 5, n=6,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day -2, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 1, predose, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 1, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 1, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 1, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 2, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 3, predose, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 3, 1 hour, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 3, 3 hour, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 3, 6 hour, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  IL-4, Session 4, Day 4, n=5,0 | 0.000 (0.0000) |
  IL-4, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 4, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 3, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 4, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 5, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day -2, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 1, predose, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 1, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 1, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 1, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 2, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 3, predose, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 3, 1 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 3, 3 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 3, 6 hour, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 4, n=4,0 | 0.000 (0.0000) |
  IL-4, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-4, Session 6, Day 5, n=4,0 | 0.000 (0.0000) |
  IL-8, Session 1, Day 1, predose, n=6,1 | 4.377 (5.8881) | 1.140 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-8, Session 1, Day 1, 1 hour, n=6,1 | 4.887 (12.0436) | 0.450 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-8, Session 1, Day 1, 3 hour, n=6,1 | 1.097 (6.7834) | 0.480 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-8, Session 1, Day 1, 6 hour, n=6,1 | 4.400 (9.5000) | 8.350 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-8, Session 1, Day 2, n=6,1 | 10.977 (25.4607) | 12.720 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-8, Session 1, Day 3, predose, n=6,1 | 6.830 (10.6309) | 9.350 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  IL-8, Session 1, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 1, Day 3, 1 hour, n=6,0 | 3.035 (6.9193) |
  IL-8, Session 1, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 1, Day 3, 3 hour, n=6,0 | -0.788 (4.9840) |
  IL-8, Session 1, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 1, Day 3, 6 hour, n=6,0 | -0.490 (7.3654) |
  IL-8, Session 1, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 1, Day 4, n=6,0 | -0.542 (5.0480) |
  IL-8, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 1, Day 5, n=6,0 | 1.198 (3.0063) |
  IL-8, Session 2, Day -2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day -2, n=6,0 | 7.848 (12.9271) |
  IL-8, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 1, predose, n=6,0 | 4.920 (8.3853) |
  IL-8, Session 2, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 1, 1 hour, n=6,0 | 1.592 (6.9965) |
  IL-8, Session 2, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 1, 3 hour, n=6,0 | 0.275 (7.2669) |
  IL-8, Session 2, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 1, 6 hour, n=6,0 | 1.243 (6.1976) |
  IL-8, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 2, n=6,0 | 5.468 (7.5652) |
  IL-8, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 3, predose, n=6,0 | 8.322 (5.0082) |
  IL-8, Session 2, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 3, 1 hour, n=6,0 | 6.432 (10.6402) |
  IL-8, Session 2, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 3, 3 hour, n=6,0 | -1.107 (5.8160) |
  IL-8, Session 2, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 3, 6 hour, n=6,0 | -0.870 (4.6278) |
  IL-8, Session 2, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 4, n=6,0 | 1.667 (5.5170) |
  IL-8, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 2, Day 5, n=6,0 | 2.853 (5.4769) |
  IL-8, Session 3, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 3, Day -2, n=5,0 | 12.742 (7.8571) |
  IL-8, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 1, predose, n=6,0 | 7.635 (6.3602) |
  IL-8, Session 3, Day 1, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 1, 1 hour, n=6,0 | 3.848 (5.5264) |
  IL-8, Session 3, Day 1, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 1, 3 hour, n=6,0 | -0.517 (5.6983) |
  IL-8, Session 3, Day 1, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 1, 6 hour, n=6,0 | 0.933 (8.0166) |
  IL-8, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 3, Day 2, n=5,0 | 3.024 (5.5819) |
  IL-8, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 3, predose, n=6,0 | 14.440 (13.4971) |
  IL-8, Session 3, Day 3, 1 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 3, 1 hour, n=6,0 | 4.887 (5.2130) |
  IL-8, Session 3, Day 3, 3 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 3, 3 hour, n=6,0 | 0.088 (4.3970) |
  IL-8, Session 3, Day 3, 6 hour, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 3, 6 hour, n=6,0 | 2.450 (6.2029) |
  IL-8, Session 3, Day 4, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 4, n=6,0 | 3.680 (4.5662) |
  IL-8, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  IL-8, Session 3, Day 5, n=6,0 | 7.783 (3.9382) |
  IL-8, Session 4, Day -2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day -2, n=5,0 | 15.686 (10.4436) |
  IL-8, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 1, predose, n=5,0 | 9.910 (11.2178) |
  IL-8, Session 4, Day 1, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 1, 1 hour, n=5,0 | 10.088 (13.7154) |
  IL-8, Session 4, Day 1, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 1, 3 hour, n=5,0 | 5.242 (11.1547) |
  IL-8, Session 4, Day 1, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 1, 6 hour, n=5,0 | 6.992 (12.0857) |
  IL-8, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 2, n=5,0 | 4.282 (8.9442) |
  IL-8, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 3, predose, n=5,0 | 15.072 (11.8360) |
  IL-8, Session 4, Day 3, 1 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 3, 1 hour, n=5,0 | 10.536 (8.8924) |
  IL-8, Session 4, Day 3, 3 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 3, 3 hour, n=5,0 | 1.474 (3.3523) |
  IL-8, Session 4, Day 3, 6 hour, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 3, 6 hour, n=5,0 | 1.208 (3.6252) |
  IL-8, Session 4, Day 4, n=5,0: number analyzed (Participants) | 5 | 0
  IL-8, Session 4, Day 4, n=5,0 | 7.118 (14.6164) |
  IL-8, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 4, Day 5, n=4,0 | -1.795 (4.8526) |
  IL-8, Session 5, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day -2, n=4,0 | 21.055 (14.5161) |
  IL-8, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 1, predose, n=4,0 | 18.213 (16.0292) |
  IL-8, Session 5, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 1, 1 hour, n=4,0 | 17.667 (15.2020) |
  IL-8, Session 5, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 1, 3 hour, n=4,0 | 12.463 (16.7548) |
  IL-8, Session 5, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 1, 6 hour, n=4,0 | 5.617 (8.7263) |
  IL-8, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 2, n=4,0 | 5.463 (9.5943) |
  IL-8, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 3, predose, n=4,0 | 16.915 (13.4207) |
  IL-8, Session 5, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 3, 1 hour, n=4,0 | 9.240 (11.0353) |
  IL-8, Session 5, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 3, 3 hour, n=4,0 | 5.902 (9.1992) |
  IL-8, Session 5, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 3, 6 hour, n=4,0 | 5.335 (7.4134) |
  IL-8, Session 5, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 4, n=4,0 | 7.610 (12.4139) |
  IL-8, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 5, Day 5, n=4,0 | 7.330 (14.2059) |
  IL-8, Session 6, Day -2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day -2, n=4,0 | 12.908 (11.2540) |
  IL-8, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 1, predose, n=4,0 | 17.575 (14.9713) |
  IL-8, Session 6, Day 1, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 1, 1 hour, n=4,0 | 18.718 (14.2024) |
  IL-8, Session 6, Day 1, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 1, 3 hour, n=4,0 | 13.823 (18.3486) |
  IL-8, Session 6, Day 1, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 1, 6 hour, n=4,0 | 12.923 (15.0125) |
  IL-8, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 2, n=4,0 | 13.338 (15.7070) |
  IL-8, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 3, predose, n=4,0 | 25.338 (17.9965) |
  IL-8, Session 6, Day 3, 1 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 3, 1 hour, n=4,0 | 11.733 (12.1142) |
  IL-8, Session 6, Day 3, 3 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 3, 3 hour, n=4,0 | 6.853 (7.9858) |
  IL-8, Session 6, Day 3, 6 hour, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 3, 6 hour, n=4,0 | 7.220 (9.8022) |
  IL-8, Session 6, Day 4, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 4, n=4,0 | 13.500 (13.0942) |
  IL-8, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  IL-8, Session 6, Day 5, n=4,0 | 14.130 (9.1046) |

21. Secondary Outcome: Change From Baseline in Fluid Phase Complement Marker-Complement 3 (C3) Over Time
Description: Blood samples were collected for assessment of Fluid Phase Complement Markers which included complement 3 (C3). Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 1 to 6: Day 1 (predose, 2,4,8 hours), Day 2, Day 3 (predose, 2,4,8 hours), Day 5, Day 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Grams per Liter (g/L)
  C3, Session 1, Day 1, predose, n=6,1 | -0.032 (0.1444) | -0.150 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  C3, Session 1, Day 1, 2 hour, n=6,1 | -0.008 (0.1105) | -0.230 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  C3, Session 1, Day 1, 4 hour, n=6,1 | 0.030 (0.0566) | -0.100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  C3, Session 1, Day 1, 8 hour, n=6,1 | 0.068 (0.2073) | -0.160 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  C3, Session 1, Day 2, n=6,1 | -0.125 (0.1033) | -0.180 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  C3, Session 1, Day 3, predose, n=6,1 | -0.198 (0.1607) | -0.200 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  C3, Session 1, Day 3, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 1, Day 3, 2 hour, n=6,0 | -0.188 (0.1572) |
  C3, Session 1, Day 3, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 1, Day 3, 4 hour, n=6,0 | -0.222 (0.1288) |
  C3, Session 1, Day 3, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 1, Day 3, 8 hour, n=6,0 | -0.155 (0.1590) |
  C3, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 1, Day 5, n=6,0 | -0.280 (0.1646) |
  C3, Session 1, Day 6, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 1, Day 6, n=6,0 | -0.338 (0.1969) |
  C3, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 1, predose, n=6,0 | -0.067 (0.1999) |
  C3, Session 2, Day 1, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 1, 2 hour, n=6,0 | -0.103 (0.1629) |
  C3, Session 2, Day 1, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 1, 4 hour, n=6,0 | -0.075 (0.2017) |
  C3, Session 2, Day 1, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 1, 8 hour, n=6,0 | -0.130 (0.1585) |
  C3, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 2, n=6,0 | -0.153 (0.1485) |
  C3, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 3, predose, n=6,0 | -0.263 (0.1385) |
  C3, Session 2, Day 3, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 3, 2 hour, n=6,0 | -0.242 (0.1694) |
  C3, Session 2, Day 3, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 3, 4 hour, n=6,0 | -0.243 (0.1994) |
  C3, Session 2, Day 3, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 3, 8 hour, n=6,0 | -0.235 (0.1685) |
  C3, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 5, n=6,0 | -0.280 (0.1716) |
  C3, Session 2, Day 6, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 2, Day 6, n=6,0 | -0.327 (0.2298) |
  C3, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 1, predose, n=6,0 | -0.053 (0.1928) |
  C3, Session 3, Day 1, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 1, 2 hour, n=6,0 | -0.078 (0.2279) |
  C3, Session 3, Day 1, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 1, 4 hour, n=6,0 | -0.058 (0.2299) |
  C3, Session 3, Day 1, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 1, 8 hour, n=6,0 | -0.057 (0.1999) |
  C3, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 3, Day 2, n=5,0 | -0.084 (0.2792) |
  C3, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 3, predose, n=6,0 | -0.215 (0.1576) |
  C3, Session 3, Day 3, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 3, 2 hour, n=6,0 | -0.232 (0.1699) |
  C3, Session 3, Day 3, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 3, 4 hour, n=6,0 | -0.200 (0.1808) |
  C3, Session 3, Day 3, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 3, 8 hour, n=6,0 | -0.190 (0.2287) |
  C3, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 5, n=6,0 | -0.290 (0.1719) |
  C3, Session 3, Day 6, n=6,0: number analyzed (Participants) | 6 | 0
  C3, Session 3, Day 6, n=6,0 | -0.308 (0.2077) |
  C3, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 1, predose, n=5,0 | -0.094 (0.2271) |
  C3, Session 4, Day 1, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 1, 2 hour, n=5,0 | -0.088 (0.1993) |
  C3, Session 4, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 4, Day 1, 4 hour, n=4,0 | -0.005 (0.1392) |
  C3, Session 4, Day 1, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 1, 8 hour, n=5,0 | -0.124 (0.1747) |
  C3, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 2, n=5,0 | -0.144 (0.1641) |
  C3, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 3, predose, n=5,0 | -0.214 (0.2454) |
  C3, Session 4, Day 3, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 3, 2 hour, n=5,0 | -0.204 (0.2306) |
  C3, Session 4, Day 3, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 3, 4 hour, n=5,0 | -0.190 (0.2088) |
  C3, Session 4, Day 3, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 3, 8 hour, n=5,0 | -0.188 (0.2305) |
  C3, Session 4, Day 5, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 5, n=5,0 | -0.270 (0.1996) |
  C3, Session 4, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  C3, Session 4, Day 6, n=5,0 | -0.302 (0.2251) |
  C3, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 1, predose, n=4,0 | -0.173 (0.1863) |
  C3, Session 5, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 1, 2 hour, n=4,0 | -0.147 (0.2326) |
  C3, Session 5, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 1, 4 hour, n=4,0 | -0.125 (0.1741) |
  C3, Session 5, Day 1, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 1, 8 hour, n=4,0 | -0.150 (0.1881) |
  C3, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 2, n=4,0 | -0.178 (0.2340) |
  C3, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 3, predose, n=4,0 | -0.248 (0.1919) |
  C3, Session 5, Day 3, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 3, 2 hour, n=4,0 | -0.235 (0.1964) |
  C3, Session 5, Day 3, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 3, 4 hour, n=4,0 | -0.280 (0.2045) |
  C3, Session 5, Day 3, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 3, 8 hour, n=4,0 | -0.235 (0.2301) |
  C3, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 5, n=4,0 | -0.258 (0.2035) |
  C3, Session 5, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 5, Day 6, n=4,0 | -0.288 (0.1941) |
  C3, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 1, predose, n=4,0 | -0.152 (0.2144) |
  C3, Session 6, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 1, 2 hour, n=4,0 | -0.145 (0.1877) |
  C3, Session 6, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 1, 4 hour, n=4,0 | -0.145 (0.2528) |
  C3, Session 6, Day 1, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 1, 8 hour, n=4,0 | -0.135 (0.2626) |
  C3, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 2, n=4,0 | -0.203 (0.2090) |
  C3, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 3, predose, n=4,0 | -0.215 (0.2319) |
  C3, Session 6, Day 3, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 3, 2 hour, n=4,0 | -0.273 (0.2179) |
  C3, Session 6, Day 3, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 3, 4 hour, n=4,0 | -0.235 (0.2243) |
  C3, Session 6, Day 3, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 3, 8 hour, n=4,0 | -0.238 (0.2421) |
  C3, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 5, n=4,0 | -0.288 (0.2269) |
  C3, Session 6, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  C3, Session 6, Day 6, n=4,0 | -0.315 (0.2225) |

22. Secondary Outcome: Change From Baseline in Fluid Phase Complement Marker-Complement 4 (C4) Over Time
Description: Blood samples were collected for assessment of Fluid Phase Complement Markers which included complement 4 (C4). Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 2, Day 5, Day 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Grams per Liter (g/L)
  C4, Session 1, Day 2, n=6,1 | -0.015 (0.0373) | 0.000 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  C4, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  C4, Session 1, Day 5, n=6,0 | -0.013 (0.0393) |
  C4, Session 1, Day 6, n=6,0: number analyzed (Participants) | 6 | 0
  C4, Session 1, Day 6, n=6,0 | -0.017 (0.0403) |
  C4, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  C4, Session 2, Day 2, n=6,0 | -0.027 (0.0423) |
  C4, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  C4, Session 2, Day 5, n=6,0 | -0.023 (0.0505) |
  C4, Session 2, Day 6, n=6,0: number analyzed (Participants) | 6 | 0
  C4, Session 2, Day 6, n=6,0 | -0.030 (0.0540) |
  C4, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  C4, Session 3, Day 2, n=5,0 | -0.010 (0.0543) |
  C4, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  C4, Session 3, Day 5, n=6,0 | -0.042 (0.0449) |
  C4, Session 3, Day 6, n=6,0: number analyzed (Participants) | 6 | 0
  C4, Session 3, Day 6, n=6,0 | -0.042 (0.0542) |
  C4, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  C4, Session 4, Day 2, n=5,0 | -0.022 (0.0531) |
  C4, Session 4, Day 5, n=5,0: number analyzed (Participants) | 5 | 0
  C4, Session 4, Day 5, n=5,0 | -0.036 (0.0677) |
  C4, Session 4, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  C4, Session 4, Day 6, n=5,0 | -0.042 (0.0507) |
  C4, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  C4, Session 5, Day 2, n=4,0 | -0.028 (0.0574) |
  C4, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  C4, Session 5, Day 5, n=4,0 | -0.033 (0.0574) |
  C4, Session 5, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  C4, Session 5, Day 6, n=4,0 | -0.025 (0.0545) |
  C4, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  C4, Session 6, Day 2, n=4,0 | -0.043 (0.0544) |
  C4, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  C4, Session 6, Day 5, n=4,0 | -0.050 (0.0678) |
  C4, Session 6, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  C4, Session 6, Day 6, n=4,0 | -0.045 (0.0666) |

23. Secondary Outcome: Change From Baseline in Fluid Phase Complement Marker-Total Complement (CH50) Over Time
Description: Blood samples were collected for assessment of Fluid Phase Complement Markers which included total complement (CH50). Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 1 to 6: Day 1 (predose, 2,4,8 hours), Day 2, Day 3 (predose, 2,4,8 hours), Day 5, Day 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units per milliliter
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Units per milliliter
  CH50, Session 1, Day 1, predose, n=6,1 | -0.7 (1.37) | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CH50, Session 1, Day 1, 2 hour, n=6,1 | -0.8 (1.33) | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CH50, Session 1, Day 1, 4 hour, n=6,1 | 0.2 (0.41) | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CH50, Session 1, Day 1, 8 hour, n=6,1 | -0.8 (1.60) | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CH50, Session 1, Day 2, n=6,1 | -2.7 (3.20) | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CH50, Session 1, Day 3, predose, n=6,1 | -3.3 (4.46) | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CH50, Session 1, Day 3, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 1, Day 3, 2 hour, n=6,0 | -3.3 (4.37) |
  CH50, Session 1, Day 3, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 1, Day 3, 4 hour, n=6,0 | -2.5 (3.78) |
  CH50, Session 1, Day 3, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 1, Day 3, 8 hour, n=6,0 | -2.2 (3.25) |
  CH50, Session 1, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 1, Day 5, n=6,0 | -4.7 (5.01) |
  CH50, Session 1, Day 6, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 1, Day 6, n=6,0 | -7.3 (6.19) |
  CH50, Session 2, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 1, predose, n=6,0 | -1.7 (3.67) |
  CH50, Session 2, Day 1, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 1, 2 hour, n=6,0 | -2.3 (4.84) |
  CH50, Session 2, Day 1, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 1, 4 hour, n=6,0 | -2.3 (4.63) |
  CH50, Session 2, Day 1, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 1, 8 hour, n=6,0 | -3.5 (7.84) |
  CH50, Session 2, Day 2, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 2, n=6,0 | -4.3 (6.02) |
  CH50, Session 2, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 3, predose, n=6,0 | -4.5 (6.16) |
  CH50, Session 2, Day 3, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 3, 2 hour, n=6,0 | -4.0 (5.55) |
  CH50, Session 2, Day 3, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 3, 4 hour, n=6,0 | -3.8 (6.31) |
  CH50, Session 2, Day 3, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 3, 8 hour, n=6,0 | -3.8 (3.92) |
  CH50, Session 2, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 5, n=6,0 | -5.2 (6.31) |
  CH50, Session 2, Day 6, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 2, Day 6, n=6,0 | -8.5 (9.61) |
  CH50, Session 3, Day 1, predose, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 1, predose, n=6,0 | -4.5 (7.94) |
  CH50, Session 3, Day 1, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 1, 2 hour, n=6,0 | -4.2 (7.44) |
  CH50, Session 3, Day 1, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 1, 4 hour, n=6,0 | -4.5 (7.79) |
  CH50, Session 3, Day 1, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 1, 8 hour, n=6,0 | -4.8 (8.35) |
  CH50, Session 3, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 3, Day 2, n=5,0 | -3.6 (8.68) |
  CH50, Session 3, Day 3, predose, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 3, predose, n=6,0 | -5.2 (8.86) |
  CH50, Session 3, Day 3, 2 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 3, 2 hour, n=6,0 | -5.2 (8.86) |
  CH50, Session 3, Day 3, 4 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 3, 4 hour, n=6,0 | -5.3 (8.57) |
  CH50, Session 3, Day 3, 8 hour, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 3, 8 hour, n=6,0 | -6.8 (10.05) |
  CH50, Session 3, Day 5, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 5, n=6,0 | -7.0 (10.28) |
  CH50, Session 3, Day 6, n=6,0: number analyzed (Participants) | 6 | 0
  CH50, Session 3, Day 6, n=6,0 | -8.2 (11.02) |
  CH50, Session 4, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 1, predose, n=5,0 | -3.0 (5.20) |
  CH50, Session 4, Day 1, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 1, 2 hour, n=5,0 | -2.0 (3.94) |
  CH50, Session 4, Day 1, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 1, 4 hour, n=5,0 | -1.6 (4.77) |
  CH50, Session 4, Day 1, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 1, 8 hour, n=5,0 | -1.6 (3.21) |
  CH50, Session 4, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 2, n=5,0 | -1.6 (3.13) |
  CH50, Session 4, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 3, predose, n=5,0 | -5.0 (6.08) |
  CH50, Session 4, Day 3, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 3, 2 hour, n=5,0 | -3.2 (4.09) |
  CH50, Session 4, Day 3, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 3, 4 hour, n=5,0 | -3.0 (6.40) |
  CH50, Session 4, Day 3, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 3, 8 hour, n=5,0 | -4.0 (6.04) |
  CH50, Session 4, Day 5, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 5, n=5,0 | -5.6 (7.70) |
  CH50, Session 4, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  CH50, Session 4, Day 6, n=5,0 | -6.6 (7.83) |
  CH50, Session 5, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 1, predose, n=4,0 | -3.8 (5.91) |
  CH50, Session 5, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 1, 2 hour, n=4,0 | -3.0 (5.72) |
  CH50, Session 5, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 1, 4 hour, n=4,0 | -2.8 (6.29) |
  CH50, Session 5, Day 1, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 1, 8 hour, n=4,0 | -3.0 (5.29) |
  CH50, Session 5, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 2, n=4,0 | -3.5 (5.32) |
  CH50, Session 5, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 3, predose, n=4,0 | -5.0 (5.77) |
  CH50, Session 5, Day 3, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 3, 2 hour, n=4,0 | -4.8 (6.80) |
  CH50, Session 5, Day 3, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 3, 4 hour, n=4,0 | -4.8 (6.70) |
  CH50, Session 5, Day 3, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 3, 8 hour, n=4,0 | -4.8 (6.80) |
  CH50, Session 5, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 5, n=4,0 | -5.5 (7.72) |
  CH50, Session 5, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 5, Day 6, n=4,0 | -5.3 (8.54) |
  CH50, Session 6, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 1, predose, n=4,0 | -2.3 (4.03) |
  CH50, Session 6, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 1, 2 hour, n=4,0 | -2.8 (6.90) |
  CH50, Session 6, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 1, 4 hour, n=4,0 | -3.3 (7.27) |
  CH50, Session 6, Day 1, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 1, 8 hour, n=4,0 | -3.5 (6.66) |
  CH50, Session 6, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 2, n=4,0 | -4.3 (6.13) |
  CH50, Session 6, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 3, predose, n=4,0 | -5.0 (8.52) |
  CH50, Session 6, Day 3, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 3, 2 hour, n=4,0 | -4.8 (8.54) |
  CH50, Session 6, Day 3, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 3, 4 hour, n=4,0 | -4.3 (8.66) |
  CH50, Session 6, Day 3, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 3, 8 hour, n=4,0 | -5.0 (8.52) |
  CH50, Session 6, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 5, n=4,0 | -5.3 (9.00) |
  CH50, Session 6, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  CH50, Session 6, Day 6, n=4,0 | -5.5 (9.47) |

24. Secondary Outcome: Change From Baseline in Inflammatory Biomarkers Over Time
Description: Blood samples were collected for assessment of inflammatory biomarkers which included C-Reactive protein (CRP), high-sensitivity C-reactive protein (hsCRP), serum amyloid A protein (SAA). Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 1 to 6: Day 1 (predose, 2,4,8 hours), Day 2, Day 3 (predose, 2,4,8 hours), Day 5, Day 6
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Milligrams per Liter (mg/L)
  CRP, Session 1, Day 1, predose, n=5,1: number analyzed (Participants) | 5 | 1
  CRP, Session 1, Day 1, predose, n=5,1 | -0.12 (0.572) | -4.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CRP, Session 1, Day 1, 2 hour, n=5,1: number analyzed (Participants) | 5 | 1
  CRP, Session 1, Day 1, 2 hour, n=5,1 | -0.26 (0.573) | -4.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CRP, Session 1, Day 1, 4 hour, n=4,1: number analyzed (Participants) | 4 | 1
  CRP, Session 1, Day 1, 4 hour, n=4,1 | -0.28 (0.486) | -4.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CRP, Session 1, Day 1, 8 hour, n=5,1: number analyzed (Participants) | 5 | 1
  CRP, Session 1, Day 1, 8 hour, n=5,1 | -0.18 (0.634) | -4.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CRP, Session 1, Day 2, n=5,1: number analyzed (Participants) | 5 | 1
  CRP, Session 1, Day 2, n=5,1 | 0.64 (1.701) | 44.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CRP, Session 1, Day 3, predose, n=5,1: number analyzed (Participants) | 5 | 1
  CRP, Session 1, Day 3, predose, n=5,1 | 14.08 (12.511) | 131.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  CRP, Session 1, Day 3, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 1, Day 3, 2 hour, n=5,0 | 14.52 (13.128) |
  CRP, Session 1, Day 3, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 1, Day 3, 4 hour, n=5,0 | 15.30 (13.119) |
  CRP, Session 1, Day 3, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 1, Day 3, 8 hour, n=5,0 | 17.64 (14.527) |
  CRP, Session 1, Day 5, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 1, Day 5, n=5,0 | 17.20 (14.772) |
  CRP, Session 1, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 1, Day 6, n=5,0 | 19.52 (15.665) |
  CRP, Session 2, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 2, Day 1, predose, n=5,0 | 2.24 (2.864) |
  CRP, Session 2, Day 1, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 2, Day 1, 2 hour, n=5,0 | 2.12 (2.613) |
  CRP, Session 2, Day 1, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 2, Day 1, 4 hour, n=5,0 | 2.18 (2.710) |
  CRP, Session 2, Day 1, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 2, Day 1, 8 hour, n=5,0 | 2.18 (2.658) |
  CRP, Session 2, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 2, Day 2, n=4,0 | 2.00 (2.624) |
  CRP, Session 2, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 2, Day 3, predose, n=5,0 | 27.42 (26.283) |
  CRP, Session 2, Day 3, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 2, Day 3, 2 hour, n=5,0 | 29.46 (27.415) |
  CRP, Session 2, Day 3, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 2, Day 3, 4 hour, n=5,0 | 30.90 (27.961) |
  CRP, Session 2, Day 3, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 2, Day 3, 8 hour, n=5,0 | 31.76 (27.897) |
  CRP, Session 2, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 2, Day 5, n=4,0 | 28.33 (22.386) |
  CRP, Session 2, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 2, Day 6, n=5,0 | 27.04 (18.632) |
  CRP, Session 3, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 1, predose, n=4,0 | 1.93 (2.343) |
  CRP, Session 3, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 1, 2 hour, n=4,0 | 2.05 (2.626) |
  CRP, Session 3, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 1, 4 hour, n=4,0 | 2.15 (2.891) |
  CRP, Session 3, Day 1, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 1, 8 hour, n=4,0 | 2.15 (2.760) |
  CRP, Session 3, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 2, n=4,0 | 1.75 (2.161) |
  CRP, Session 3, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 3, predose, n=4,0 | 18.13 (15.476) |
  CRP, Session 3, Day 3, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 3, 2 hour, n=4,0 | 19.40 (16.403) |
  CRP, Session 3, Day 3, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 3, 4 hour, n=4,0 | 21.20 (17.827) |
  CRP, Session 3, Day 3, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 3, 8 hour, n=4,0 | 22.63 (18.466) |
  CRP, Session 3, Day 5, n=5,0: number analyzed (Participants) | 5 | 0
  CRP, Session 3, Day 5, n=5,0 | 19.00 (15.625) |
  CRP, Session 3, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 3, Day 6, n=4,0 | 24.10 (16.785) |
  CRP, Session 4, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 1, predose, n=4,0 | 2.33 (4.487) |
  CRP, Session 4, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 1, 2 hour, n=4,0 | 2.53 (4.762) |
  CRP, Session 4, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 1, 4 hour, n=4,0 | 2.45 (4.669) |
  CRP, Session 4, Day 1, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 1, 8 hour, n=4,0 | 2.40 (4.455) |
  CRP, Session 4, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 2, n=4,0 | 2.23 (3.963) |
  CRP, Session 4, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 3, predose, n=4,0 | 12.45 (13.533) |
  CRP, Session 4, Day 3, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 3, 2 hour, n=4,0 | 14.75 (16.539) |
  CRP, Session 4, Day 3, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 3, 4 hour, n=4,0 | 16.75 (19.129) |
  CRP, Session 4, Day 3, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 3, 8 hour, n=4,0 | 17.30 (17.830) |
  CRP, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 5, n=4,0 | 18.43 (9.959) |
  CRP, Session 4, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  CRP, Session 4, Day 6, n=4,0 | 19.98 (11.277) |
  CRP, Session 5, Day 1, predose, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 5, Day 1, predose, n=3,0 | 2.23 (3.439) |
  CRP, Session 5, Day 1, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 5, Day 1, 2 hour, n=3,0 | 2.13 (3.350) |
  CRP, Session 5, Day 1, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 5, Day 1, 4 hour, n=3,0 | 1.97 (3.147) |
  CRP, Session 5, Day 1, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 5, Day 1, 8 hour, n=3,0 | 2.10 (3.378) |
  CRP, Session 5, Day 2, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 5, Day 2, n=3,0 | 1.37 (2.811) |
  CRP, Session 5, Day 3, predose, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 5, Day 3, predose, n=3,0 | 8.33 (11.517) |
  CRP, Session 5, Day 3, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 5, Day 3, 2 hour, n=3,0 | 9.87 (12.881) |
  CRP, Session 5, Day 3, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 5, Day 3, 4 hour, n=3,0 | 10.47 (12.874) |
  CRP, Session 5, Day 3, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 5, Day 3, 8 hour, n=3,0 | 12.90 (14.944) |
  CRP, Session 5, Day 5, n=2,0: number analyzed (Participants) | 2 | 0
  CRP, Session 5, Day 5, n=2,0 | 34.30 (40.588) |
  CRP, Session 5, Day 6, n=2,0: number analyzed (Participants) | 2 | 0
  CRP, Session 5, Day 6, n=2,0 | 35.20 (34.931) |
  CRP, Session 6, Day 1, predose, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 1, predose, n=3,0 | 4.00 (3.851) |
  CRP, Session 6, Day 1, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 1, 2 hour, n=3,0 | 3.63 (3.711) |
  CRP, Session 6, Day 1, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 1, 4 hour, n=3,0 | 3.70 (3.835) |
  CRP, Session 6, Day 1, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 1, 8 hour, n=3,0 | 3.70 (3.874) |
  CRP, Session 6, Day 2, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 2, n=3,0 | 2.63 (2.914) |
  CRP, Session 6, Day 3, predose, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 3, predose, n=3,0 | 9.17 (8.879) |
  CRP, Session 6, Day 3, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 3, 2 hour, n=3,0 | 11.10 (10.887) |
  CRP, Session 6, Day 3, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 3, 4 hour, n=3,0 | 12.70 (11.555) |
  CRP, Session 6, Day 3, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 3, 8 hour, n=3,0 | 14.67 (12.580) |
  CRP, Session 6, Day 5, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 5, n=3,0 | 14.10 (7.146) |
  CRP, Session 6, Day 6, n=3,0: number analyzed (Participants) | 3 | 0
  CRP, Session 6, Day 6, n=3,0 | 17.33 (7.844) |
  hsCRP, Session 1, Day 1, predose, n=5,1: number analyzed (Participants) | 5 | 1
  hsCRP, Session 1, Day 1, predose, n=5,1 | -0.08 (0.356) | -3.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  hsCRP, Session 1, Day 1, 2 hour, n=5,1: number analyzed (Participants) | 5 | 1
  hsCRP, Session 1, Day 1, 2 hour, n=5,1 | -0.08 (0.327) | -3.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  hsCRP, Session 1, Day 1, 4 hour, n=4,1: number analyzed (Participants) | 4 | 1
  hsCRP, Session 1, Day 1, 4 hour, n=4,1 | -0.20 (0.271) | -3.70 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  hsCRP, Session 1, Day 1, 8 hour, n=5,1: number analyzed (Participants) | 5 | 1
  hsCRP, Session 1, Day 1, 8 hour, n=5,1 | -0.10 (0.406) | -3.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  hsCRP, Session 1, Day 2, n=5,1: number analyzed (Participants) | 5 | 1
  hsCRP, Session 1, Day 2, n=5,1 | 0.56 (1.286) | 41.40 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  hsCRP, Session 1, Day 3, predose, n=5,1: number analyzed (Participants) | 5 | 1
  hsCRP, Session 1, Day 3, predose, n=5,1 | 14.54 (13.149) | 135.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  hsCRP, Session 1, Day 3, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 1, Day 3, 2 hour, n=5,0 | 15.14 (13.363) |
  hsCRP, Session 1, Day 3, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 1, Day 3, 4 hour, n=5,0 | 15.84 (13.607) |
  hsCRP, Session 1, Day 3, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 1, Day 3, 8 hour, n=5,0 | 17.10 (14.294) |
  hsCRP, Session 1, Day 5, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 1, Day 5, n=5,0 | 16.70 (14.332) |
  hsCRP, Session 1, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 1, Day 6, n=5,0 | 18.60 (14.778) |
  hsCRP, Session 2, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 2, Day 1, predose, n=5,0 | 1.88 (2.539) |
  hsCRP, Session 2, Day 1, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 2, Day 1, 2 hour, n=5,0 | 1.78 (2.351) |
  hsCRP, Session 2, Day 1, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 2, Day 1, 4 hour, n=5,0 | 1.90 (2.478) |
  hsCRP, Session 2, Day 1, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 2, Day 1, 8 hour, n=5,0 | 1.78 (2.179) |
  hsCRP, Session 2, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 2, Day 2, n=4,0 | 1.75 (2.266) |
  hsCRP, Session 2, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 2, Day 3, predose, n=5,0 | 26.76 (26.122) |
  hsCRP, Session 2, Day 3, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 2, Day 3, 2 hour, n=5,0 | 29.28 (27.373) |
  hsCRP, Session 2, Day 3, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 2, Day 3, 4 hour, n=5,0 | 30.36 (27.018) |
  hsCRP, Session 2, Day 3, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 2, Day 3, 8 hour, n=5,0 | 31.10 (26.885) |
  hsCRP, Session 2, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 2, Day 5, n=4,0 | 28.13 (21.919) |
  hsCRP, Session 2, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  hsCRP, Session 2, Day 6, n=5,0 | 27.20 (18.468) |
  hsCRP, Session 3, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 1, predose, n=4,0 | 1.60 (2.017) |
  hsCRP, Session 3, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 1, 2 hour, n=4,0 | 1.63 (2.175) |
  hsCRP, Session 3, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 1, 4 hour, n=4,0 | 1.70 (2.403) |
  hsCRP, Session 3, Day 1, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 1, 8 hour, n=4,0 | 1.65 (2.161) |
  hsCRP, Session 3, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 2, n=4,0 | 1.25 (1.754) |
  hsCRP, Session 3, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 3, predose, n=4,0 | 17.88 (15.954) |
  hsCRP, Session 3, Day 3, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 3, 2 hour, n=4,0 | 19.23 (16.675) |
  hsCRP, Session 3, Day 3, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 3, 4 hour, n=4,0 | 20.58 (17.733) |
  hsCRP, Session 3, Day 3, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 3, 8 hour, n=4,0 | 22.10 (18.149) |
  hsCRP, Session 3, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 5, n=4,0 | 22.45 (15.042) |
  hsCRP, Session 3, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 3, Day 6, n=4,0 | 23.73 (16.141) |
  hsCRP, Session 4, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 1, predose, n=4,0 | 2.28 (4.043) |
  hsCRP, Session 4, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 1, 2 hour, n=4,0 | 2.53 (4.610) |
  hsCRP, Session 4, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 1, 4 hour, n=4,0 | 2.53 (4.479) |
  hsCRP, Session 4, Day 1, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 1, 8 hour, n=4,0 | 2.58 (4.528) |
  hsCRP, Session 4, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 2, n=4,0 | 2.20 (3.558) |
  hsCRP, Session 4, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 3, predose, n=4,0 | 12.33 (13.881) |
  hsCRP, Session 4, Day 3, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 3, 2 hour, n=4,0 | 14.40 (16.324) |
  hsCRP, Session 4, Day 3, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 3, 4 hour, n=4,0 | 16.00 (18.240) |
  hsCRP, Session 4, Day 3, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 3, 8 hour, n=4,0 | 17.08 (17.972) |
  hsCRP, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 5, n=4,0 | 19.60 (10.903) |
  hsCRP, Session 4, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  hsCRP, Session 4, Day 6, n=4,0 | 20.73 (11.391) |
  hsCRP, Session 5, Day 1, predose, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 5, Day 1, predose, n=3,0 | 2.03 (3.349) |
  hsCRP, Session 5, Day 1, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 5, Day 1, 2 hour, n=3,0 | 1.97 (3.320) |
  hsCRP, Session 5, Day 1, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 5, Day 1, 4 hour, n=3,0 | 1.83 (3.175) |
  hsCRP, Session 5, Day 1, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 5, Day 1, 8 hour, n=3,0 | 1.87 (3.323) |
  hsCRP, Session 5, Day 2, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 5, Day 2, n=3,0 | 1.23 (2.574) |
  hsCRP, Session 5, Day 3, predose, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 5, Day 3, predose, n=3,0 | 9.10 (13.182) |
  hsCRP, Session 5, Day 3, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 5, Day 3, 2 hour, n=3,0 | 10.43 (14.629) |
  hsCRP, Session 5, Day 3, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 5, Day 3, 4 hour, n=3,0 | 11.17 (14.865) |
  hsCRP, Session 5, Day 3, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 5, Day 3, 8 hour, n=3,0 | 12.67 (15.557) |
  hsCRP, Session 5, Day 5, n=2,0: number analyzed (Participants) | 2 | 0
  hsCRP, Session 5, Day 5, n=2,0 | 33.95 (40.941) |
  hsCRP, Session 5, Day 6, n=2,0: number analyzed (Participants) | 2 | 0
  hsCRP, Session 5, Day 6, n=2,0 | 34.80 (34.083) |
  hsCRP, Session 6, Day 1, predose, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 1, predose, n=3,0 | 3.77 (3.853) |
  hsCRP, Session 6, Day 1, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 1, 2 hour, n=3,0 | 3.37 (3.523) |
  hsCRP, Session 6, Day 1, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 1, 4 hour, n=3,0 | 3.50 (3.799) |
  hsCRP, Session 6, Day 1, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 1, 8 hour, n=3,0 | 3.27 (3.584) |
  hsCRP, Session 6, Day 2, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 2, n=3,0 | 2.33 (2.775) |
  hsCRP, Session 6, Day 3, predose, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 3, predose, n=3,0 | 8.97 (9.752) |
  hsCRP, Session 6, Day 3, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 3, 2 hour, n=3,0 | 10.57 (11.075) |
  hsCRP, Session 6, Day 3, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 3, 4 hour, n=3,0 | 12.60 (12.322) |
  hsCRP, Session 6, Day 3, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 3, 8 hour, n=3,0 | 15.33 (14.276) |
  hsCRP, Session 6, Day 5, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 5, n=3,0 | 14.43 (7.801) |
  hsCRP, Session 6, Day 6, n=3,0: number analyzed (Participants) | 3 | 0
  hsCRP, Session 6, Day 6, n=3,0 | 18.63 (8.607) |
  SAA, Session 1, Day 1, predose, n=5,1: number analyzed (Participants) | 5 | 1
  SAA, Session 1, Day 1, predose, n=5,1 | 0.2164 (1.55486) | -22.3723 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  SAA, Session 1, Day 1, 2 hour, n=5,1: number analyzed (Participants) | 5 | 1
  SAA, Session 1, Day 1, 2 hour, n=5,1 | 0.1738 (1.13909) | -22.4187 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  SAA, Session 1, Day 1, 4 hour, n=5,1: number analyzed (Participants) | 5 | 1
  SAA, Session 1, Day 1, 4 hour, n=5,1 | 0.3902 (1.56253) | -21.7463 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  SAA, Session 1, Day 1, 8 hour, n=5,1: number analyzed (Participants) | 5 | 1
  SAA, Session 1, Day 1, 8 hour, n=5,1 | 0.2695 (1.57992) | -14.8767 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  SAA, Session 1, Day 2, n=5,1: number analyzed (Participants) | 5 | 1
  SAA, Session 1, Day 2, n=5,1 | 2.9247 (3.47577) | 322.2895 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  SAA, Session 1, Day 3, predose, n=5,1: number analyzed (Participants) | 5 | 1
  SAA, Session 1, Day 3, predose, n=5,1 | 50.7137 (55.02969) | 1437.7667 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  SAA, Session 1, Day 3, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 1, Day 3, 2 hour, n=5,0 | 54.8466 (59.36005) |
  SAA, Session 1, Day 3, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 1, Day 3, 4 hour, n=5,0 | 54.9329 (55.92645) |
  SAA, Session 1, Day 3, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 1, Day 3, 8 hour, n=5,0 | 68.4699 (75.51138) |
  SAA, Session 1, Day 5, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 1, Day 5, n=5,0 | 54.6741 (69.66316) |
  SAA, Session 1, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 1, Day 6, n=5,0 | 55.2882 (63.77870) |
  SAA, Session 2, Day 1, predose, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 1, predose, n=5,0 | 1.0277 (1.64965) |
  SAA, Session 2, Day 1, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 1, 2 hour, n=5,0 | 0.9841 (2.22042) |
  SAA, Session 2, Day 1, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 1, 4 hour, n=5,0 | 1.4543 (2.61184) |
  SAA, Session 2, Day 1, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 1, 8 hour, n=5,0 | 1.0588 (1.52455) |
  SAA, Session 2, Day 2, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 2, n=5,0 | 3.7244 (1.63856) |
  SAA, Session 2, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 3, predose, n=5,0 | 134.4489 (160.14208) |
  SAA, Session 2, Day 3, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 3, 2 hour, n=5,0 | 145.2507 (171.92591) |
  SAA, Session 2, Day 3, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 3, 4 hour, n=5,0 | 142.5438 (174.11156) |
  SAA, Session 2, Day 3, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 3, 8 hour, n=5,0 | 100.8836 (184.35963) |
  SAA, Session 2, Day 5, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 5, n=5,0 | 76.8593 (136.83379) |
  SAA, Session 2, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 2, Day 6, n=5,0 | 101.0688 (105.88787) |
  SAA, Session 3, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 3, Day 1, predose, n=4,0 | 0.2428 (1.13002) |
  SAA, Session 3, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 3, Day 1, 2 hour, n=4,0 | 0.1863 (1.06333) |
  SAA, Session 3, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 3, Day 1, 4 hour, n=4,0 | 0.0475 (1.00422) |
  SAA, Session 3, Day 1, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 3, Day 1, 8 hour, n=5,0 | 4.0339 (8.62955) |
  SAA, Session 3, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 3, Day 2, n=4,0 | 6.4822 (11.14119) |
  SAA, Session 3, Day 3, predose, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 3, Day 3, predose, n=5,0 | 54.7393 (82.22346) |
  SAA, Session 3, Day 3, 2 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 3, Day 3, 2 hour, n=5,0 | 58.0526 (83.12677) |
  SAA, Session 3, Day 3, 4 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 3, Day 3, 4 hour, n=5,0 | 64.1995 (93.61736) |
  SAA, Session 3, Day 3, 8 hour, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 3, Day 3, 8 hour, n=5,0 | 66.9605 (93.98658) |
  SAA, Session 3, Day 5, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 3, Day 5, n=5,0 | 58.6742 (50.93398) |
  SAA, Session 3, Day 6, n=5,0: number analyzed (Participants) | 5 | 0
  SAA, Session 3, Day 6, n=5,0 | 49.4029 (46.30012) |
  SAA, Session 4, Day 1, predose, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 1, predose, n=4,0 | -0.1305 (1.86822) |
  SAA, Session 4, Day 1, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 1, 2 hour, n=4,0 | 0.0159 (1.91086) |
  SAA, Session 4, Day 1, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 1, 4 hour, n=4,0 | -0.0013 (1.84104) |
  SAA, Session 4, Day 1, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 1, 8 hour, n=4,0 | 0.1997 (1.70496) |
  SAA, Session 4, Day 2, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 2, n=4,0 | 1.6015 (1.07082) |
  SAA, Session 4, Day 3, predose, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 3, predose, n=4,0 | 45.1067 (82.67535) |
  SAA, Session 4, Day 3, 2 hour, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 3, 2 hour, n=4,0 | 51.0650 (94.33211) |
  SAA, Session 4, Day 3, 4 hour, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 3, 4 hour, n=4,0 | 55.0009 (101.37965) |
  SAA, Session 4, Day 3, 8 hour, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 3, 8 hour, n=4,0 | 55.7135 (101.39069) |
  SAA, Session 4, Day 5, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 5, n=4,0 | 51.2002 (54.84780) |
  SAA, Session 4, Day 6, n=4,0: number analyzed (Participants) | 4 | 0
  SAA, Session 4, Day 6, n=4,0 | 41.2457 (38.77052) |
  SAA, Session 5, Day 1, predose, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 1, predose, n=3,0 | -0.1498 (1.04561) |
  SAA, Session 5, Day 1, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 1, 2 hour, n=3,0 | -0.2399 (0.89843) |
  SAA, Session 5, Day 1, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 1, 4 hour, n=3,0 | -0.1906 (0.94124) |
  SAA, Session 5, Day 1, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 1, 8 hour, n=3,0 | -0.1771 (0.95814) |
  SAA, Session 5, Day 2, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 2, n=3,0 | 0.1380 (0.61958) |
  SAA, Session 5, Day 3, predose, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 3, predose, n=3,0 | 10.8884 (17.72052) |
  SAA, Session 5, Day 3, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 3, 2 hour, n=3,0 | 8.6783 (11.48176) |
  SAA, Session 5, Day 3, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 3, 4 hour, n=3,0 | 9.2527 (11.23663) |
  SAA, Session 5, Day 3, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 3, 8 hour, n=3,0 | 13.7941 (19.39827) |
  SAA, Session 5, Day 5, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 5, n=3,0 | 66.2542 (107.98594) |
  SAA, Session 5, Day 6, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 5, Day 6, n=3,0 | 73.0823 (118.07036) |
  SAA, Session 6, Day 1, predose, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 1, predose, n=3,0 | 1.2964 (1.75482) |
  SAA, Session 6, Day 1, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 1, 2 hour, n=3,0 | 1.0538 (1.74392) |
  SAA, Session 6, Day 1, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 1, 4 hour, n=3,0 | 1.3139 (2.18542) |
  SAA, Session 6, Day 1, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 1, 8 hour, n=3,0 | 0.9078 (1.72500) |
  SAA, Session 6, Day 2, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 2, n=3,0 | 1.2641 (0.89837) |
  SAA, Session 6, Day 3, predose, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 3, predose, n=3,0 | 7.4697 (5.41886) |
  SAA, Session 6, Day 3, 2 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 3, 2 hour, n=3,0 | 8.3574 (4.40865) |
  SAA, Session 6, Day 3, 4 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 3, 4 hour, n=3,0 | 11.0305 (8.80978) |
  SAA, Session 6, Day 3, 8 hour, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 3, 8 hour, n=3,0 | 14.5333 (12.26460) |
  SAA, Session 6, Day 5, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 5, n=3,0 | 25.2529 (27.55204) |
  SAA, Session 6, Day 6, n=3,0: number analyzed (Participants) | 3 | 0
  SAA, Session 6, Day 6, n=3,0 | 32.6318 (41.82856) |

25. Secondary Outcome: Maximum Concentration (Cmax) of GSK2398852
Description: Blood samples were collected for evaluation of Pharmacokinetic (PK) parameters including Cmax at indicated time points. Geometric mean and geometric coefficient of variation of Cmax is presented.
Time Frame: Session 1 to 6: Day 1 (Pre-dose, 6, 8, 12 hour), Day 2, Day 3 (Pre-dose and at 6 hour), Day 4, Day 7 and Day 11
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (ug/mL)
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Micrograms per milliliter (ug/mL)
  Session 1, n=6,1 | 86.94 (31.58) | 88.64 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed.
  Session 2, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, n=6,0 | 235.48 (25.22) |
  Session 3, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, n=6,0 | 222.23 (44.40) |
  Session 4, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, n=5,0 | 179.82 (33.87) |
  Session 5, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, n=4,0 | 185.52 (34.06) |
  Session 6, n=4,0: number analyzed (Participants) | 4 | 0
  Session 6, n=4,0 | 228.51 (49.73) |

26. Secondary Outcome: Time Associated With Cmax (Tmax) of GSK2398852
Description: Blood samples were collected for evaluation of PK parameters including Tmax at indicated time points. Median and full range of Tmax is presented.
Time Frame: Session 1 to 6: Day 1 (Pre-dose, 6, 8, 12 hour), Day 2, Day 3 (Pre-dose and at 6 hour), Day 4, Day 7 and Day 11
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Hour
  Session 1, n=6,1 | 54.18 [53.9 to 54.9] | 6.1 [6.1 to 6.1]
  Session 2, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, n=6,0 | 54.07 [53.3 to 54.7] |
  Session 3, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, n=6,0 | 54.06 [12.1 to 55.8] |
  Session 4, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, n=5,0 | 54.50 [53.9 to 56.1] |
  Session 5, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, n=4,0 | 54.28 [6.1 to 56.1] |
  Session 6, n=4,0: number analyzed (Participants) | 4 | 0
  Session 6, n=4,0 | 54.18 [53.9 to 56.0] |

27. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time t (AUC 0-t) of GSK2398852
Description: Blood samples were collected for evaluation of PK parameters including AUC 0-t at indicated time points. Geometric mean and geometric coefficient of variation of AUC0-t is presented.
Time Frame: Session 1 to 6: Day 1 (Pre-dose, 6, 8, 12 hour), Day 2, Day 3 (Pre-dose and at 6 hour), Day 4, Day 7 and Day 11
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter (h*ug/mL)
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Hour*micrograms per milliliter (h*ug/mL)
  Session 1, n=6,1 | 5130.0 (46.72) | 2148.2 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, n=6,0 | 14610.1 (34.73) |
  Session 3, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, n=6,0 | 13804.6 (50.34) |
  Session 4, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, n=5,0 | 12970.9 (51.52) |
  Session 5, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, n=4,0 | 15595.3 (51.13) |
  Session 6, n=4,0: number analyzed (Participants) | 4 | 0
  Session 6, n=4,0 | 17126.7 (43.98) |

28. Secondary Outcome: Cmax of GSK2315698 for Newly Diagnosed Mayo Stage II/IIIa AL Amyloidosis Participants
Description: Blood samples were planned to be collected for evaluation of PK parameters including Cmax at indicated time points for GSK2315698 for newly diagnosed Mayo stage II/IIIa AL Amyloidosis participants. However, no participant was enrolled in 'Group 3: Newly diagnosed Mayo stage II/IIIa AL participants.'
Time Frame: Day 1: Pre-dose; Day 2 (pre-dose and 2 hours post-dose); Day 3: Pre-dose in each session (each session of 24 days)
Population: Safety Population. Data was not collected for this outcome due to blood samples were not collected to evaluate PK of GSK2315698 as no participant was enrolled in 'Group 3: Newly diagnosed Mayo stage II/IIIa AL participants'.
Arm/Group | Group 3: Newly Diagnosed Mayo Stage II/IIIa AL Participants
Number analyzed (Participants) | 0

29. Secondary Outcome: Tmax of GSK2315698 for Newly Diagnosed Mayo Stage II/IIIa AL Amyloidosis Participants
Description: Blood samples were planned to be collected for evaluation of PK parameters including Tmax at indicated time points for GSK2315698 for newly diagnosed Mayo stage II/IIIa AL Amyloidosis participants. However, no participant was enrolled in 'Group 3: Newly diagnosed Mayo stage II/IIIa AL participants'.
Time Frame: Day 1: Pre-dose; Day 2: pre-dose and 2 hours post-dose; Day 3: Pre-dose in each session (each session of 24 days)
Population: as for outcome 28
Arm/Group | Group 3: Newly Diagnosed Mayo Stage II/IIIa AL Participants
Number analyzed (Participants) | 0

30. Secondary Outcome: AUC 0-t of GSK2315698 for Newly Diagnosed Mayo Stage II/IIIa AL Amyloidosis Participants
Description: Blood samples were planned to be collected for evaluation of PK parameters including AUC0-t at indicated time points for GSK2315698 for newly diagnosed Mayo stage II/IIIa AL Amyloidosis participants. However, no participant was enrolled in 'Group 3: Newly diagnosed Mayo stage II/IIIa AL participants'.
Time Frame: Day 1: Pre-dose; Day 2 (pre-dose and 2 hours post-dose); Day 3: Pre-dose in each session (each session of 24 days)
Population: as for outcome 28
Arm/Group | Group 3: Newly Diagnosed Mayo Stage II/IIIa AL Participants
Number analyzed (Participants) | 0

31. Secondary Outcome: Change From Baseline in Global Longitudinal Strain (GLS) by CMR
Description: Global Longitudinal Strain was measured by CMR at indicated time points. GLS included feature tracking and tagging by CMR. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 2 to 5: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of myocardial shortening
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Percentage of myocardial shortening
  GLS Tagging, Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  GLS Tagging, Session 2, Day 24, n=6,0 | 0.003 (0.2907) |
  GLS Tagging, Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  GLS Tagging, Session 3, Day 24, n=6,0 | 0.229 (0.5836) |
  GLS Tagging, Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  GLS Tagging, Session 4, Day 24, n=5,0 | 0.392 (0.4121) |
  GLS Tagging, Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  GLS Tagging, Session 5, Day 24, n=4,0 | 0.349 (0.9354) |
  GLS Tagging, 8 Week follow-up, n=6,1 | 1.125 (1.6448) | -3.404 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  GLS Tagging, 6 month follow-up, n=2,0: number analyzed (Participants) | 2 | 0
  GLS Tagging, 6 month follow-up, n=2,0 | -1.014 (0.3654) |
  GLS Feature Tracking, Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  GLS Feature Tracking, Session 2, Day 24, n=6,0 | 1.729 (2.3613) |
  GLS Feature Tracking, Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  GLS Feature Tracking, Session 3, Day 24, n=6,0 | 0.803 (2.3712) |
  GLS Feature Tracking, Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  GLS Feature Tracking, Session 4, Day 24, n=5,0 | 1.326 (4.0639) |
  GLS Feature Tracking, Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  GLS Feature Tracking, Session 5, Day 24, n=4,0 | 1.657 (2.1277) |
  GLS Feature Tracking, 8 Week follow-up, n=6,1 | 0.639 (1.3678) | 3.951 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  GLS Feature Tracking, 6 month follow-up, n=2,0: number analyzed (Participants) | 2 | 0
  GLS Feature Tracking, 6 month follow-up, n=2,0 | 1.234 (4.6888) |

32. Secondary Outcome: Change From Baseline in GLS by ECHO
Description: Global Longitudinal Strain was measured by ECHO at indicated time points. GLS included speckle tracking by ECHO. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 1 to 6: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of myocardial shortening
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Percentage of myocardial shortening
  GLS Speckle Tracking, Session 1, Day 24, n=6,1 | -3.55 (5.709) | -0.90 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  GLS Speckle Tracking, Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  GLS Speckle Tracking, Session 2, Day 24, n=6,0 | -0.58 (6.013) |
  GLS Speckle Tracking, Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  GLS Speckle Tracking, Session 3, Day 24, n=6,0 | -1.17 (7.487) |
  GLS Speckle Tracking, Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  GLS Speckle Tracking, Session 4, Day 24, n=5,0 | 1.26 (5.299) |
  GLS Speckle Tracking, Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  GLS Speckle Tracking, Session 5, Day 24, n=4,0 | 1.13 (9.044) |
  GLS Speckle Tracking, Session 6, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  GLS Speckle Tracking, Session 6, Day 24, n=4,0 | -2.08 (4.555) |
  GLS Speckle Tracking, 8 Week follow-up, n=6,1 | -1.82 (10.013) | 1.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  GLS Speckle Tracking, 6 month follow-up, n=4,0: number analyzed (Participants) | 4 | 0
  GLS Speckle Tracking, 6 month follow-up, n=4,0 | 0.40 (4.268) |

33. Secondary Outcome: Change From Baseline in LV Twist Over Time
Description: LV twist was measured by CMR at indicated time points. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 2 to 5: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Degree
  Session 2, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  Session 2, Day 24, n=5,0 | 0.550 (1.6672) |
  Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, Day 24, n=6,0 | 0.431 (2.4369) |
  Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, Day 24, n=5,0 | -0.611 (1.8979) |
  Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, Day 24, n=4,0 | -0.628 (1.2269) |
  8 Week follow-up, n=6,1 | -0.264 (2.0835) | 0.914 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  6 month follow-up, n=2,0: number analyzed (Participants) | 2 | 0
  6 month follow-up, n=2,0 | -0.633 (0.3349) |

34. Secondary Outcome: Change From Baseline in Stroke Volume (SV) by CMR
Description: Stroke volume is the amount of blood ejected by the left ventricle in one contraction. SV was measured by CMR at indicated time points. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 2 to 5: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Milliliter
  Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, Day 24, n=6,0 | -2.760 (7.8305) |
  Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, Day 24, n=6,0 | -1.228 (24.3834) |
  Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, Day 24, n=5,0 | -9.766 (9.7838) |
  Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, Day 24, n=4,0 | -11.477 (14.4238) |
  8 Week follow-up, n=6,1 | 2.400 (19.1252) | -6.750 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  6 month follow-up, n=2,0: number analyzed (Participants) | 2 | 0
  6 month follow-up, n=2,0 | -6.160 (12.0491) |

35. Secondary Outcome: Change From Baseline in SV by ECHO
Description: Stroke volume is the amount of blood ejected by the left ventricle in one contraction. SV was measured by ECHO at indicated time points. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 1 to 6: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Milliliter
  Session 1, Day 24, n=6,1 | 2.580 (5.4518) | -5.640 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, Day 24, n=6,0 | -1.885 (4.6569) |
  Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, Day 24, n=6,0 | -1.398 (8.0106) |
  Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, Day 24, n=5,0 | -7.484 (6.5228) |
  Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, Day 24, n=4,0 | -9.043 (9.5173) |
  Session 6, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 6, Day 24, n=4,0 | -5.095 (7.1431) |
  8 Week follow-up, n=6,1 | -4.343 (7.3457) | -6.490 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  6 month follow-up, n=4,0: number analyzed (Participants) | 4 | 0
  6 month follow-up, n=4,0 | -4.275 (9.9743) |

36. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (EF) by CMR
Description: Left ventricular ejection fraction is a measurement of the percentage of blood leaving the heart each time it contracts. EF was measured by CMR at indicated time points. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 2 to 5: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of ejected blood
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Percentage of ejected blood
  Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, Day 24, n=6,0 | 0.100 (3.9071) |
  Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, Day 24, n=6,0 | 0.687 (11.7171) |
  Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, Day 24, n=5,0 | -3.380 (5.4750) |
  Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, Day 24, n=4,0 | -3.257 (7.9513) |
  8 Week follow-up, n=6,1 | -1.258 (7.9932) | -2.800 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  6 month follow-up, n=2,0: number analyzed (Participants) | 2 | 0
  6 month follow-up, n=2,0 | 0.680 (8.7681) |

37. Secondary Outcome: Change From Baseline in Left Ventricular EF by ECHO
Description: Left ventricular ejection fraction is a measurement of the percentage of blood leaving the heart each time it contracts. EF was measured by ECHO at indicated time points. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 1 to 6: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of ejected blood
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Percentage of ejected blood
  Session 1, Day 24, n=6,1 | 2.10 (5.707) | -7.40 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, Day 24, n=6,0 | -0.38 (3.111) |
  Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, Day 24, n=6,0 | -0.30 (3.318) |
  Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, Day 24, n=5,0 | -2.74 (5.766) |
  Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, Day 24, n=4,0 | -4.05 (7.832) |
  Session 6, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 6, Day 24, n=4,0 | -3.53 (3.288) |
  8 Week follow-up, n=6,1 | -1.72 (8.471) | -3.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  6 month follow-up, n=4,0: number analyzed (Participants) | 4 | 0
  6 month follow-up, n=4,0 | 1.20 (3.442) |

38. Secondary Outcome: Change From Baseline in Left Ventricle End Diastolic Volume (EDV) by CMR
Description: Left ventricle EDV is the volume of blood in the left ventricle at end load or filling in (diastole) or the amount of blood in the ventricles just before systole. EDV was measured by CMR at indicated time points. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 2 to 5: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Milliliter
  Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, Day 24, n=6,0 | -3.473 (11.2584) |
  Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, Day 24, n=6,0 | 1.653 (7.3322) |
  Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, Day 24, n=5,0 | -5.262 (5.3765) |
  Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, Day 24, n=4,0 | -9.323 (11.5275) |
  8 Week follow-up, n=6,1 | 9.887 (19.3925) | -4.560 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  6 month follow-up, n=2,0: number analyzed (Participants) | 2 | 0
  6 month follow-up, n=2,0 | -21.030 (8.0469) |

39. Secondary Outcome: Change From Baseline in Left Ventricle End Diastolic Volume (EDV) by ECHO
Description: Left ventricle EDV is the volume of blood in the left ventricle at end load or filling in (diastole) or the amount of blood in the ventricles just before systole. EDV was measured by ECHO at indicated time points. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 1 to 6: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Milliliter
  Session 1, Day 24, n=6,1 | 0.050 (4.6276) | -1.790 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 2, Day 24, n=6,0 | -2.940 (10.2320) |
  Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  Session 3, Day 24, n=6,0 | -2.922 (14.0019) |
  Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  Session 4, Day 24, n=5,0 | -12.338 (10.2249) |
  Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 5, Day 24, n=4,0 | -11.860 (14.5676) |
  Session 6, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  Session 6, Day 24, n=4,0 | -5.073 (11.3679) |
  8 Week follow-up, n=6,1 | -7.648 (4.4630) | -7.100 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  6 month follow-up, n=4,0: number analyzed (Participants) | 4 | 0
  6 month follow-up, n=4,0 | -12.045 (20.2972) |

40. Secondary Outcome: Change From Baseline in Ratio of Mitral Peak Velocity of Early Filling to Early Diastolic Mitral Annual Velocity (E/e' Ratio)
Description: E/e' ratio was measured by ECHO at indicated time points. It had 2 separate measurements: lateral and septal. Baseline was considered as the latest assessment prior to first administration of either study drug, i.e. CPHPC or anti-SAP mAb. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Session 1 to 6: Day 24; 8 week follow-up; 6 months follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
Number analyzed (Participants) | 6 | 1
Ratio
  E/e Lateral Ratio, Session 1, Day 24, n=6,1 | -1.55 (2.813) | -2.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  E/e Lateral Ratio, Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  E/e Lateral Ratio, Session 2, Day 24, n=6,0 | -0.77 (3.555) |
  E/e Lateral Ratio, Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  E/e Lateral Ratio, Session 3, Day 24, n=6,0 | 3.20 (2.197) |
  E/e Lateral Ratio, Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  E/e Lateral Ratio, Session 4, Day 24, n=5,0 | -0.64 (4.750) |
  E/e Lateral Ratio, Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  E/e Lateral Ratio, Session 5, Day 24, n=4,0 | 1.22 (5.134) |
  E/e Lateral Ratio, Session 6, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  E/e Lateral Ratio, Session 6, Day 24, n=4,0 | 3.25 (2.300) |
  E/e Lateral Ratio, 8 Week follow-up, n=6,1 | 0.05 (2.681) | 2.90 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  E/e Lateral Ratio, 6 month follow-up, n=4,0: number analyzed (Participants) | 4 | 0
  E/e Lateral Ratio, 6 month follow-up, n=4,0 | -0.58 (4.442) |
  E/e Septal Ratio, Session 1, Day 24, n=6,1 | 0.50 (2.995) | -2.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  E/e Septal Ratio, Session 2, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  E/e Septal Ratio, Session 2, Day 24, n=6,0 | 0.52 (4.640) |
  E/e Septal Ratio, Session 3, Day 24, n=6,0: number analyzed (Participants) | 6 | 0
  E/e Septal Ratio, Session 3, Day 24, n=6,0 | 5.33 (5.136) |
  E/e Septal Ratio, Session 4, Day 24, n=5,0: number analyzed (Participants) | 5 | 0
  E/e Septal Ratio, Session 4, Day 24, n=5,0 | 2.96 (3.462) |
  E/e Septal Ratio, Session 5, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  E/e Septal Ratio, Session 5, Day 24, n=4,0 | 4.48 (3.010) |
  E/e Septal Ratio, Session 6, Day 24, n=4,0: number analyzed (Participants) | 4 | 0
  E/e Septal Ratio, Session 6, Day 24, n=4,0 | 6.23 (5.917) |
  E/e Septal Ratio, 8 Week follow-up, n=6,0: number analyzed (Participants) | 6 | 0
  E/e Septal Ratio, 8 Week follow-up, n=6,0 | 2.83 (4.236) |
  E/e Septal Ratio, 6 month follow-up, n=4,0: number analyzed (Participants) | 4 | 0
  E/e Septal Ratio, 6 month follow-up, n=4,0 | 4.95 (1.708) |

ADVERSE EVENTS:
Time Frame: Non-serious AEs were collected from start of study treatment (Week 0) up to 56 days after the last dosing session (up to 265 days). SAEs were collected from start of the study treatment (Week 0) up to the end of study (Up to 369 days).
Description: SAEs and non-serious AEs are reported for Safety Population for Group 1 and 2 only as no participant was enrolled in Group-3.
Arm/Group | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants | Group 2: Post-chemotherapy AL Amyloidosis Participants
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/1
Other Adverse Events (participants affected / at risk) | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants (N=6) | Group 2: Post-chemotherapy AL Amyloidosis Participants (N=1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Cardiac TTR Amyloidosis (ATTR-CM) Participants (N=6) | Group 2: Post-chemotherapy AL Amyloidosis Participants (N=1)
Constipation (Gastrointestinal disorders) | 3 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 3 (6) | 1 (1)
Fatigue (General disorders) | 3 (9) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Catheter site dermatitis (General disorders) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Secretion discharge (General disorders) | 1 (2) | 0 (0)
Thirst (General disorders) | 1 (2) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Somnolence (Nervous system disorders) | 2 (8) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (33) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 3 (12) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (2) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Urine output increased (Investigations) | 1 (1) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03044353/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT03044353/SAP_001.pdf